## **Effects of Code Sepsis Implementation on ED Sepsis Care (Code Sepsis)**

**Protocol version:** Version 9.0

**Updated:** February 1, 2023

Principal Investigator: Ithan Peltan, MD, MSc

**Trial steering committee:** Ithan Peltan, MD, MSc

Samuel Brown, MD, MPH Joseph Bledsoe, MD

Facilities involved: Intermountain Medical Center

**Utah Valley Hospital** 

Dixie Regional Medical Center

**Sponsor:** National Institutes of Health (1K23 GM12966-01A1)

## TABLE OF CONTENTS

| 1. | . ABBREVIATIONS AND DEFINITIONS | 4 |
|---|---|---|
| | 1.1 Abbreviations | 4 |
| | 1.2 Definitions | 5 |
| 2. | STUDY SUMMARY | 6 |
| | 2.1 Title | 6 |
| | 2.2 Primary Objective | 6 |
| | 2.3 Primary Hypothesis | 6 |
| | 2.4 Study Design | 6 |
| | 2.4.1 Study groups and phases | 6 |
| | 2.4.2 Inclusion criteria | |
| | 2.4.3 Exclusion criteria | |
| | 2.4.5 Primary analysis cohort | |
| | 2.4.6 Primary outcome | |
| | 2.4.7 Secondary outcomes | |
| | 2.4.9 Sample size | |
| 2 | TRIAL DESCRIPTION | |
| J. | 3.1 Background | |
| | 3.2 Overall Study Motivation, Aim and Hypothesis | |
| | 3.3 Primary Objective | |
| | 3.4 Primary Hypothesis | |
| | 3.5 Study Overview | |
| | 3.6 Analysis cohorts | |
| | 3.6.1 Primary analysis cohort | |
| | 3.6.2 Secondary and sensitivity analysis cohorts | |
| | 3.6.3 Subgroups | |
| | 3.7 Endpoints | 10 |
| | 3.7.1 Primary outcome | 10 |
| | 3.7.2 Secondary outcomes | |
| 4. | STUDY POPULATION AND ENROLLMENT | 12 |
| | 4.1 Setting | 12 |
| | 4.2 Study Population | |
| | 4.2.1 Exposure groups | |
| | 4.2.2 Inclusion criteria: | |
| | 4.2.3 Exclusion criteria: | |
| | 4.2.4 Inclusion/exclusion criteria rationale | |
| | 4.3 Waivers of Informed Consent and HIPAA authorization | |
| | 4.4 Minorities and Women | |
| _ | 4.5 Vulnerable Subjects | |
| 5. | STUDY PROCEDURES | |
| | 5.1 Standard Care | |
| | 5.2 Code Sepsis Protocol | |
| 6. | DATA COLLECTION AND VARIABLES | |
| | 6.1 Data Collection | |
| | 6.2 Anonymous Data Collection For Protocol Development and During Live Code Sepsis Activa | |
| | 6.3 Active Follow-I In for Patients Lindergoing Code Sensis | 18<br>18 |
| | N ⊀ //CTIVE FOUNW-LIN FOR POTIENTS LINGERGOING ( ORE SENSIS | 1 12 |

| | 6.4 Protected Health Information | 18 |
|---|---|---|
| | 6.5 Variables/data elements | 18 |
| | 6.6 Data Management | 20 |
| 7. | DATA ANALYSIS | 21 |
| | 7.1 Introduction to Quasi-Experimental Analysis | |
| | 7.2 Multivariable models | |
| | 7.3 Sample size/power analysis | |
| 0 | RISK ASSESSMENT | |
| ο. | 8.1 Potential Risks | |
| | 8.1.1 Risk of confidentiality breach | |
| | 8.1.2 Risks for control group patients | |
| | 8.1.3. Risks to patients exposed to the Code Sepsis protocol | |
| | 8.2 Alternatives to Participation | |
| | 8.3 Minimization of Risks | |
| | 8.3.1 Protections against invasion of privacy or breach of confidentiality | |
| | 8.3.2 Incidental findings | |
| | 8.3.3 Protection against medicolegal risk | |
| | 8.3.4 Optimization of Code Sepsis targeting | |
| | 8.3.4 Protections against overtreatment and anchoring bias | |
| | 8.3.5 Protections against overtreatment and adverse drug reactions | |
| | 8.4 Potential Benefits of the Proposed Research to Human Subjects and Others | |
| | 8.5 Importance of the Knowledge to be Gained | |
| a | HUMAN SUBJECTS | |
| ٦. | 9.1 Selection of Subjects | |
| | 9.2 Waiver of Informed Consent and HIPAA Authorization | |
| | 9.2.1 Research involves no more than minimal risk | |
| | 9.2.2 No adverse effects on the rights and welfare of participants | |
| | 9.2.3 The research could not practicably be carried out without waiver of informed consent | |
| | 9.2.4 Information on the Code Sepsis protocol and study will be available to all ED patients | |
| | 9.2.5 The minimal necessary amount of protected information will be obtained | |
| | 9.2.6 All data, including PHI, will be securely guarded from improper disclosure | |
| 10 | ). MONITORING AND SAFETY REPORTING | 28 |
| | 10.1 Potential Risks and Benefits for Participants | 28 |
| | 10.2 Adverse Event and Serious Adverse Event Collection | |
| | 10.2.1 Adverse event | 28 |
| | 10.2.2 Serious Adverse Event (SAE) | |
| | 10.2.3 Adverse event monitoring | |
| | 10.3 Adverse Event and Serious Adverse Event Reporting | 29 |
| | 10.4 Interim Analysis | 30 |
| | 10.5 Data and Safety Monitoring | |
| | 10.5.1 Safety Monitoring Procedures | 30 |
| | 10.5.2 Enrollment, procedure, regulatory, and data quality monitoring | 31 |
| | 10.5.3 Frequency of data and safety monitoring | |
| | 10.5.4 Independent safety monitor identify and affiliation | |
| | 10.5.5 Conflict of interest for independent safety monitor | |
| | 10.5.6 Independent safety monitor responsibilities | |
| | 10.6 Confidentiality During Adverse Event Reporting | |
| | L BIBLIOGRAPHY | |
| Αl | PPENDIX A — Eligible IV and IV-equivalent antibiotics | 35 |

| APPENDIX B — "Sepsis mimic" ICD codes | 37 |
|---------------------------------------------------------|----|
| B.1 Heart failure diagnosis codes <sup>1</sup> | 37 |
| B.2 Pulmonary embolism diagnosis codes <sup>1,2</sup> | 38 |
| B.3 Deep vein thrombosis diagnosis codes <sup>1,2</sup> | 39 |
| APPENDIX C — Diagnosis codes for adverse drug reaction | |

## 1. ABBREVIATIONS AND DEFINITIONS

### 1.1 Abbreviations

**AE** = Adverse event

**CHF** = Congestive heart failure

**ED** = Emergency Department

**GCS** = Glasgow Coma Scale

HIPAA = Health Insurance Portability and Accountability Act

**IRB** = Institutional Review Board

**ICU** = Intensive Care Unit

**ICD-9-CM** = International Classification of Disease, version 9, clinical modification

**ICD-10-CM** = International Classification of Disease, version 10, clinical modification

**INR** = International normalized ratio

ISM = Independent safety monitor

ITT = Intent to treat

MAP = Mean arterial pressure

**NIH** = National Institutes of Health

**PE** = Pulmonary embolism

**PI** = Principle investigator

**PHI** = Protected Health Information

**REDCap** = Research Electronic Data Capture

**RR** = Respiratory rate

**SOFA score** = Sequential Organ Failure Assessment score

**SBP** = Systolic blood pressure

**SpO2** = Oxygen saturation via pulse oximetry

**SUSAR =** Serious and Unexpected Suspected Adverse Reactions

**SAEs=** Serious Adverse Events

WBC = White blood cell count

#### 1.2 Definitions

- Adverse Event: Any untoward medical occurrence associated with the use of a drug or a study procedure, whether or not considered drug related.
- Adverse reaction: An adverse reaction means any adverse event caused by a study intervention. An adverse reaction is a subset of all suspected adverse reactions where there is a reason to conclude that the study intervention caused the event.
- **Door-to-antibiotic time**: Primary outcome; the time from the first recorded arrival time in ED (usually ED triage or registration) and the time the first eligible antibiotic was administered.
- **Hypotension**: SBP <90 mmHg or MAP <65 mmHg or, where applicable, receipt of vasopressor medication
- Intention to Treat (ITT): All eligible patients who present to the ED will be included in the ITT cohort for the purposes of analyzing the primary and secondary study outcomes.
- **PHI:** identifiable health information that is used, maintained, stored, or transmitted by a HIPAA-covered entity
- **SAEs:** Serious Adverse Events Adverse events that are serious and unexpected and have a reasonable possibility that the event was due to a study procedure
- Sepsis: Life-threatening organ dysfunction resulting from a dysregulated host response to infection, clinically identified in the emergency department (ED) by an acute rise in the Sequential Organ Failure Assessment (SOFA) score while in the ED ≥2 points above baseline <u>plus</u> suspected or confirmed infection in the ED.1
- **Sepsis mimic:** Clinical condition which may cause patient to exhibit and/or be treated for sepsis even though infection is not actually present. For the present study, pulmonary embolism (PE) and congestive heart failure (CHF) have been identified as sepsis mimic conditions.
- Septic shock: Sepsis associated with hypotension requiring administration of vasopressors.
- Study hospital: Defined as the hospital where the patient presented to the ED.
- Suspected adverse reaction: any adverse event for which there is a reasonable possibility that the study procedures caused the adverse event. Reasonable possibility means there is evidence to suggest a causal relationship between the study procedures and the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than adverse reaction (21 CFR 312.32(a)).
- Suspected or confirmed infection in the emergency department: Identified based on clinical behaviors of clinicians as the combination of administration of an IV- or IV-equivalent antibiotic plus collection of a body fluid culture or a positive molecular test for infection.
- Suspected Unexpected Serious Adverse Reaction (SUSAR) An adverse reaction that is both
  unexpected (not consistent with the risks outlined in the protocol or investigator brochure), serious,
  and meets the definition of a Suspected Adverse Reaction

## 2. STUDY SUMMARY

### 2.1 Title

Effects of Code Sepsis Implementation on ED Sepsis Care (Code Sepsis)

## 2.2 Primary Objective

Determine the effects of reorganizing ED sepsis care (Code Sepsis protocol) on door-to-antibiotic time for ED patients with sepsis.

## 2.3 Primary Hypothesis

Early activation of a multidisciplinary, coordinated, team-based assessment and treatment protocol for patients with potential sepsis will decrease door-to-antibiotic time for ED patients with sepsis.

## 2.4 Study Design

Pragmatic phase 2a pre/post single-center implementation study with contemporaneous controls testing reorganization of standard ED sepsis care around a protocol for early, coordinated, multidisciplinary protocol for assessment of patients with potential sepsis (Code Sepsis protocol).

- 1. We will emphasize pragmatic, real-world implementation of the Code Sepsis protocol in a single ED.
- 2. We will compare care delivered to ED patients after Code Sepsis protocol implementation in the intervention ED to care received in this ED prior to Code Sepsis implementation.
- 3. We will conduct a quasi-experimental analysis using contemporaneous control data obtained from two non-intervention hospitals to control for temporal trends in studied outcomes not resulting from the tested intervention.
- 4. We will measure the effects of protocol implementation on all ED patients with sepsis (including patients not treated under the Code Sepsis protocol) as well as potential bystander effects.

## 2.4.1 Study groups and phases

Phase #1: Pre intervention (November 13, 2018 to November 12, 2019)

- Control EDs: Standard care
- Intervention ED: Standard care

Phase #2: Intervention roll-in (November 13, 2019 to February 12, 2020)

- Control EDs: Standard care
- Intervention ED: Launch and fine-tuning of Code Sepsis protocol, fine tuning of Code Sepsis activation mechanism.

Phase #3: Full intervention (February 13, 2020 to February 12, 2021)

- Control EDs: Standard care
- Intervention ED: Full implementation of Code Sepsis protocol

#### 2.4.2 Inclusion criteria

- 1. Age ≥18 years
- 2. Arrival to intervention or a control ED during study period

#### 2.4.3 Exclusion criteria

1. Age <18 years

#### 2. Trauma patient

### 2.4.5 Primary analysis cohort

ED patients with clinical sepsis, as identified by the combination of

- 1) Acute organ failure: SOFA score while in the ED ≥2 points above baseline
- 2) Suspected or confirmed infection while in the ED, as identified by both:
  - a) Administration of ≥1 IV or IV-equivalent antibiotics while in the ED
  - b) Collection of ≥1 body fluid cultures while in the ED

#### 2.4.6 Primary outcome

Door-to-antibiotic time

#### 2.4.7 Secondary outcomes

- Mortality (including 30-day, 1-year, hospital)
- Hospital charges
- Hospital length of stay
- Code Sepsis activation rate
- Code Sepsis activation accuracy
- Antibiotic utilization fraction
- Antibiotic spectrum
- Antibiotic overtreatment rate
- Adverse drug & allergic reaction incidence (e.g. anaphylaxis, new onset Clostridium difficile infection)

#### 2.4.8 Data analysis

The primary analysis will use quasi-experimental methods to compare sepsis patients' adjusted mean door-to-antibiotic time (primary outcome) at the intervention hospital pre- versus post-implementation of the Code Sepsis protocol using the measured change at non-intervention hospitals to control for preversus post-intervention changes not attributable to protocol implementation. Secondary analyses will compare the change in secondary outcomes using similar methods.

#### 2.4.9 Sample size

Assuming 4.5 sepsis patients per day at the intervention ED, treatment of 30% of these patients by Code Sepsis teams during study phase #3, and 6 total sepsis patients daily in control EDs (all conservative estimates), I will have 90% power to detect a change ≥16 minutes in the overall average door-to-antibiotic time among all ED sepsis patients after Code Sepsis implementation at the intervention hospital.

## 3. TRIAL DESCRIPTION

## 3.1 Background

Sepsis, the combination of infection and acute organ dysfunction, is a common, morbid, and often lethal syndrome. <sup>1,2</sup> Sepsis hospitalizes 1.3 million patients each year, kills 20%, and costs \$23.7 billion. <sup>2-4</sup> Early, appropriate antibiotic initiation is critical: sepsis survival decreases with every hour's delay. <sup>5-13</sup> While guidelines and government mandates thus emphasize prompt antibiotics, international guidelines' have admitted a lack of data to support the feasibility or implementation of their one-hour door-to-antibiotic goal. <sup>14,15</sup>

Among patients presenting to the emergency department (ED) with sepsis, we previously found that non-patient contextual cues could improve rapid antibiotic initiation, whereas ED busyness was associated with delayed antibiotics. <sup>16,17</sup> I also discovered five-fold variation between physicians in median door-to-antibiotic time. <sup>5</sup> ED care reorganization could bypass these cognitive, stylistic, and resource barriers to timely sepsis treatment. In fact, ED protocols linking prehospital notification to a multidisciplinary, team-based response are common and effective for trauma, stroke, and myocardial infarction, <sup>18-22</sup> conditions that are less common and less mortal than sepsis but require similarly time-sensitive treatment. <sup>23</sup> Given that sepsis has a less definitive presentation, however, analogous protocols for sepsis could waste resources or promote anchoring bias and overtreatment of patients without sepsis, issues observed with door-to-antibiotic standards for pneumonia. <sup>24-26</sup>

We hypothesize that reorganizing ED sepsis care around multidisciplinary "Code Sepsis" teams activated prior to or upon patients' ED arrival will reduce door-to-antibiotic times — with tolerable overtreatment rates — by mobilizing personnel, systematizing illness severity and infection risk assessment, <sup>27</sup> facilitating test completion, and eliminating any gap between treatment decision and antibiotic infusion. This study will therefore evaluate the effectiveness and tradeoffs of a Code Sepsis program for ED sepsis patients.

## 3.2 Overall Study Motivation, Aim and Hypothesis

Many emergency department (ED) patients with sepsis do not receive antibiotics and other care within intervals recommended in international guidelines. Efforts to accelerate treatment, however, may lead to overtreatment and other adverse effects. The goal of this project is to determine the potential effectiveness and tradeoffs of a Code Sepsis program for ED sepsis patients.

## <u>Aim</u>: Establish the feasibility and effects of a team-based Code Sepsis protocol designed to accelerate antibiotic initiation for ED patients with suspected sepsis.

Using preexisting infrastructure, implement prehospital- or triage-activated Code Sepsis ED teams in a single ED and compare sepsis patients' door-to-antibiotic times pre- and post-implementation, controlling for unrelated temporal trends with observational data from two non-intervention EDs.

<u>Hypothesis</u>: Prehospital or triage-based activation of an ED team prepared to rapidly diagnose and treat sepsis decreases door-to-antibiotic time without increasing overtreatment.

## 3.3 Primary Objective

Determine the effect of reorganizing ED sepsis care (Code Sepsis protocol) on door-to-antibiotic time for ED patients with sepsis.

## 3.4 Primary Hypothesis

Early activation of a multidisciplinary, coordinated, team-based assessment and treatment protocol for patients with potential sepsis will decrease door-to-antibiotic times for ED patients with sepsis.

## 3.5 Study Overview

To assess feasibility and test the preliminary efficacy of ED-based Code Sepsis teams activated on or before patients' ED arrival, we will pursue a Phase 2a implementation trial involving Code Sepsis team activation in one ED (Intermountain Medical Center [IMC]) while collecting contemporaneous control data at two other urban EDs (Utah Valley Hospital and Dixie Regional Medical Center [control sites], Table 1).

• Months 1-12: Collect baseline data (all sites), refine Code Sepsis protocol, and train ED staff at IMC.

Portions of baseline data may be collected in a retrospective fashion. At the intervention site during this period, we may also undertake preparatory work to Code Sepsis protocol launch, including anonymous patient care observations to evaluate care processes; pilot testing of the draft Code Sepsis protocol or its components; and testing of the



Figure 1. Code Sepsis implementation and data collection for Aim III.

accuracy of Code Sepsis activation mechanisms.

- Months 13-15: Run-in period: implement Code Sepsis protocol at IMC, optimize protocol & its trigger.
- Months 25-36: Continue Code Sepsis protocol at site A (intervention ED). Continue standard care
  processes for sepsis without change (control condition) at two non-intervention EDs

Using contemporaneous controls and rigorous statistical methods, we will assess how implementation of the Code Sepsis protocol affects process and patient outcomes in the intervention ED (Figure 1). Continuation of the Code Sepsis protocol (with or without revision) by the intervention ED and/or adoption elsewhere within the Intermountain Healthcare system is expected to be contingent on the results of these analyses.

## 3.6 Analysis cohorts

## 3.6.1 Primary analysis cohort

ED patients with clinical sepsis, as identified by the combination of

- 1) Acute organ failure: SOFA score while in the ED ≥2 points above baseline
- 2) Suspected or confirmed infection while in the ED, as identified by both:
  - c) Administration of ≥1 IV or IV-equivalent antibiotics while in the ED (see Appendix A)
  - d) Collection of ≥1 body fluid cultures while in the ED

## 3.6.2 Secondary and sensitivity analysis cohorts

- 1) All eligible ED patients
- 2) ED patients with a "sepsis mimic" diagnosis based on a primary ICD-10 discharge diagnosis codes for congestive heart failure or venous thromboembolism with no diagnostic code for infection (see Appendix B).
- 3) "Likely" sepsis patients based on simple triage assessment to include fever and at least 1 out of 3 of hypotension (SBP <90 mmHg), altered mental status (GCS ≤14), or respiratory failure (RR ≥22 or SpO2 ≤85%).

#### 3.6.3 Subgroups

A priori subgroups will include: sex; hypotension (SBP <90 mmHg or MAP <65 mmHg) present on ED arrival.

## 3.7 Endpoints

Analysis will be conducted on an intention to treat basis.

#### 3.7.1 Primary outcome

Door-to-antibiotic time among all ED sepsis patients. Door-to-antibiotic time is the time from the first recorded arrival time in ED (usually ED triage or registration) and the time the first eligible antibiotic was administered (Appendix A).

### 3.7.2 Secondary outcomes

- Clinical/patient-centered secondary outcomes (measured among all ED sepsis patients):
  - 1) All-cause mortality to day 30
  - 2) All-cause mortality to 1 year
  - 3) In-hospital all-cause mortality
  - 4) Hospital charges: Amount charged to patient for their medical care during index ED visit and associated hospitalization.
  - 5) Hospital length of stay
- Process/feasibility secondary outcomes
  - 1) Code Sepsis activation rate: Measured as the percentage of all ED patients for whom the Code Sepsis protocol was activated.
  - 2) Code Sepsis activation accuracy metrics. Accurate Code Sepsis activation is defined as activation for patients who have sepsis while in the ED and no activation for patients who do not have sepsis in the ED.
- Adverse effects and unintended outcomes of protocol implementation

- 1) Antibiotic utilization percentage: measured as the fraction of (1) all ED patients; (2) Code Sepsis activation patients; or (3) "likely" sepsis patients who received IV or IV-equivalent antibiotics.
- 2) Antibiotic spectrum: Total Stenehjem antibiotic spectrum score<sup>28</sup> for all antibiotics administered in first 24 hours, measured for (1) all ED patients or (2) sepsis patients
- 3) Antibiotic overtreatment rate: Percentage of "sepsis mimic" patients who received IV or IVequivalent antibiotics in the ED.
- 4) New onset C. difficile colitis incidence: Percentage of (1) all ED patients and (2) ED sepsis patients with a positive stool test for *Clostridium difficile* colitis between 72 hours and 90 days after ED arrival.
- 5) Adverse drug & allergic reaction incidence: Measured as the fraction of 1) all ED patients and (2) ED sepsis patients with a discharge diagnosis code consistent with anaphylaxis or with an adverse reaction to antibiotics (see Appendix C).

#### Potential exploratory outcomes

- Measures of organ failure trajectory, to include change in the SOFA score between hospital day 1 and hospital day 3, and overall and organ-specific measures of organ failure-free days through day 28.
  - Organ-failure free days (OFFD) are defined as the number of days from the time of the first SOFA score ≤1 above baseline to day 28 after ED arrival, assuming survival for at least two consecutive calendar days after the SOFA score ≤1 above baseline and continued SOFA score ≤1 point above baseline to day 28. If a patient has SOFA score rise again to ≥2 points above baseline and subsequently achieves SOFA score ≤1 point above baseline to day 28, VFDs will be counted from the end of the last period of SOFA score ≤1 to day 28. If a patient had SOFA score ≥2 points above baseline at day 27 or dies prior to day 28, OFFD will be zero
  - Support-free days (i.e. ventilator-free days) are calculated similar to OFFD
- 2) Mortality at other intervals
- 3) Testing and treatment utilization. Outcomes measured among (1) among all ED sepsis patients; (2) all ED patients; (3) "likely" sepsis patients
- 4) Code Sepsis care process timing: measured among patients who received Code Sepsis protocol activation as time from protocol activation until completion of key protocol steps, to include blood culture collection, chest X-ray collection, team huddle, antibiotic initiation
- 5) Timing of testing & care processes among all sepsis patients, to include ED clinician assessment, ED room placement, ED departure, blood culture collection, radiology testing, and order entry for antibiotics. Measured analogous to door-to-antibiotic time.
- 6) Code Sepsis protocol adherence: measured as performance of protocol steps in correct order both individually and as a fraction of all possible.

## 4. STUDY POPULATION AND ENROLLMENT

## 4.1 Setting

Intermountain Healthcare (hereafter "Intermountain") is a nonprofit health system based in Salt Lake City, Utah with 23 hospitals in Utah and Idaho. Code Sepsis implementation will occur in a teaching ED (IMC, my "home" hospital) providing 89,000 visits annually (2.8% with clinical sepsis) for an economically and ethnically diverse population of 1.1 million in Salt Lake County, Utah plus referrals

from Wyoming, Nevada, and Idaho. To avoid spillover effects, concurrent control data will be electronically abstracted from two Intermountain EDs (Utah Valley Hospital and Dixie Regional Medical Center) staffed by other physician groups (Table 1).

**Table 1.** Study hospital characteristics

| Site | Description | Hospital beds | ED<br>beds | Annual ED visits |
|---|---|---|---|---|
| IMC | Tertiary/teaching | 472 | 56 | 89,000 |
| <b>Utah Valley</b> | Regional referral | 395 | 28 | 49,000 |
| DRMC | Regional referral | 321 | 35 | 65,000 |

## 4.2 Study Population

We will study adult, non-trauma patients from the IMC ED and two control EDs during three phases (Figure 1): baseline (1 year, standard care at all sites); run-in (3 months, IMC ED launches/fine tunes the Code Sepsis protocol); and Code Sepsis implementation (1 year, Code Sepsis at IMC, standard care in control EDs). For this pre/post implementation trial, in which there will be no direct patient contact and in which we are comparing current standard care processes to a new, redesigned standard care

processes in a non-randomized fashion, all ED patients who meet inclusion and do not meet exclusion criteria will be included in the analysis.

#### 4.2.1 Exposure groups

N=135,000)

The group within which patient is analyzed is determined by the combination of (1) when the patient presents to the ED and (2) which hospital/ED to which the patient presents (Figures 1 and 2).

A. Pre-implementation control group at non-intervention hospitals: Admission to ED at nonintervention hospitals (Utah Valley



Figure 2. Subject allocation by study phase and hospital Hospital and Dixie Regional Medical Center) prior to Code Sepsis implementation (estimated

- B. Pre-implementation control group at intervention hospital: Admission to ED at IMC prior to Code Sepsis implementation (estimated N=100,000)
- C. Post-implementation control group at non-intervention hospitals: Admission to ED at nonintervention hospitals (Utah Valley Hospital and Dixie Regional Medical Center) after implementation of Code Sepsis protocol at IMC (estimated N=170,000)
- D. Exposure group: Admission to ED at IMC during full Code Sepsis implementation (estimated N=125,000)

#### 4.2.2 Inclusion criteria:

- o ED patient at Intermountain Medical Center, Utah Valley Hospital, Dixie Regional Medical Center
- ED arrival beginning 1 year prior to date of Code Sepsis implementation at Intermountain
   Medical Center and continuing through 15 months after Code Sepsis implementation date.
- Age ≥18 years

### 4.2.3 Exclusion criteria:

- Age <18 years</li>
- o Trauma patient

## 4.2.4 Inclusion/exclusion criteria rationale

Patients <18 years of age are excluded because the mechanisms, manifestations, and management of sepsis in children <18 years of age are often distinct from those applicable to adults, and in fact will vary depending on age group across childhood. Additionally, children are managed in most EDs by a distinct team of clinicians using distinct protocols. As such, prehospital or triage-based sepsis prediction models applicable to adults are unlikely to work for children <18 years. Due to the above issues, implementation of a single sepsis care protocol for individuals age <18 years and age ≥18 years would impair the efficacy, feasibility, and generalizability of the proposed Code Sepsis protocol. Trauma patients are excluded because clinical identification of these patients is straightforward and triggers preexisting team-based care protocols with options for prehospital activation.

#### 4.2.5 Study phase dates

ED patients arriving to study EDs will be assigned to a study phase based on their ED arrival date.

- Phase #1 (pre-intervention analysis phase): November 13, 2018 to November 12, 2019
- Phase #2 (intervention roll-in): November 13, 2019 to February 12, 2020
- Phase #3 (full intervention analysis phase): February 13, 2020 to February 12, 2021

### 4.3 Waivers of Informed Consent and HIPAA authorization

This study comparing standard care to a new form of standard care will be carried out under a waiver of informed consent and HIPAA authorization (see section 9).

#### 4.4 Minorities and Women

Women and minorities will be enrolled in proportion to their representation in the population base from which this study was developed, specifically patients presenting to Intermountain hospitals located in Utah's Salt Lake, Washington, and Weber Counties. In order to provide generalizable data for the ED patient diagnosis groups studied in each Aim, there will be no specific selection criteria that differ between sex/gender and racial/ethnic groups. Hospitals in this study serve counties with a combined population of over 1.5 million individuals, including over 26% who are Hispanic or non-white race. We expect the sex, ethnic and racial mix of the enrolled patients to reflect the population served.

### 4.5 Vulnerable Subjects

We anticipate that potentially vulnerable subjects are eligible for the study. Potentially vulnerable patient subjects include pregnant women, prisoners, and/or individuals with decisional impairment. The purpose of this project is to identify a cohort that reflects the diversity of the U.S. sepsis population. Therefore, we believe these individuals should not be excluded from the study since the study is of no more than minimal risk.

- 1. Data on vulnerable population membership will not be explicitly collected, and in fact attempting to identify and exclude members of potentially vulnerable populations could increase risk to both vulnerable patients and the overall subject cohort.
- 2. Altered mental status is also a common manifestation or complication of sepsis. Excluding patients with decisional impairment would therefore severely bias results of the planned analyses.
- 3. In implementation studies such as this, it is generally not possible to exclude vulnerable subjects. Aim III's intervention involves testing a new option for standard care for ED sepsis management, so excluding vulnerable populations could actually subject these patients to harm because exclusion would prevent their receiving standard care. Assessment for vulnerability status, moreover, would largely preclude the planned intervention by preventing activation of prehospital or ED triage alerts.

## 5. STUDY PROCEDURES

This study will measure the effect of a redesign of standard care for ED sepsis patients, specifically implementation of Code Sepsis protocol at Intermountain Medical Center. The study will include three phases with two groups during each phase. The primary analysis will only use data from phases #1 and #3 (see Figure 1 and 2).

<u>Phase #0:</u> Protocol development (1 year, overlaps with phase #1)

- Control EDs: N/A
- Intervention ED: A small number of suspected sepsis patients (<10) may undergo
  anonymous observation to understand care processes involved in ED sepsis care. In
  addition, testing and iterative optimization of the accuracy of the Code Sepsis activation
  may employ direct observation of care for a convenience sample of patients during ED
  triage and comparison of activation criteria to clinician judgment, final sepsis diagnosis
  based on chart review, and electronic sepsis queries. Finally, pilot testing of the draft
  protocol may be conducted on a small convenience sample of patients (<20) identified by ED
  clinicians as having possible sepsis. We will collect anonymous data about completion of
  Code Sepsis processes during pilot testing.</li>

Phase #1: Pre intervention (1 year)

- Control EDs: Standard care
- Intervention ED: Standard care.

Phase #2: Intervention roll-in

- Control EDs: Standard care
- Intervention ED: Launch and fine-tuning of Code Sepsis protocol, fine tuning of Code Sepsis activation mechanism.

Phase #3: Full intervention

- Control EDs: Standard care
- Intervention ED: Full implementation of Code Sepsis protocol

<u>Phase #4 (operational)</u>: Continuation of the Code Sepsis protocol (with or without revision) by the intervention ED and/or adoption elsewhere within the Intermountain Healthcare system is expected to be contingent on observed effects of protocol implementation. It is possible that an inadequate benefit/risk ratio could lead to a decision not to continue the Code Sepsis protocol.

#### 5.1 Standard Care

Patients arriving to the control EDs (all study phases) and the intervention ED during study Phase #1 will receive care as per then-current ED practices and protocols, guided by clinician judgment within a system-wide care process model for sepsis. As of early 2019, ED standard care for sepsis applicable at all study sites includes a standardized Care Process Model, expected completion of a standardized checklist, and standardized order sets.

## 5.2 Code Sepsis Protocol

The Code Sepsis protocol (Figure 3) has six steps developed in collaboration with ED-based study team members and ED leaders (including physicians, nurses, pharmacists, and others) from the implementation ED and the Intermountain system. The current draft protocol was further iteratively revised based on input derived from the proposed multidisciplinary team during *in situ* high-fidelity simulation and during informal/ad hoc operationally-oriented pilot testing of steps 1-5 during live patient care. The below protocol will be adapted further prior to and after implementation to ensure the protocol is feasible, efficient, and functions as intended based on stakeholder input and, as needed, additional protocol element testing during simulation and/or live patient care. Further revision will occur, during the protocol run-in phase and as needed based on observed findings and stakeholder input.



Figure 3. Current Code Sepsis protocol based on iterative revision using simulation testing, stakeholder input, & live pilot testing.

- 1) Identify likely sepsis patient from prehospital notification call data (nurse), at ED triage (nurse/physician), or on ED room placement (nurse or physician), adapting local and national practice for stroke team activation.<sup>29,30</sup>
- 2) Mobilize ED personnel and equipment to meet patients on arrival to the ED room using methods and communication networks already developed for ED trauma and stroke teams.
- 3) Concurrent patient evaluation and data collection by multiple disciplines (20-25 minutes), to include bedside assessment (e.g. history, examination, vital signs, allergy and medication history) by the physician, nurse and pharmacist; IV placement; blood and urine sampling; point-of-care laboratory testing, including lactate and urinalysis; and portable X-ray imaging. Appropriate therapeutic interventions will continue in parallel during the nominal data collection phase.
- 4) Team "huddles" to decide if sepsis diagnosis has been confirmed, disproven, or remains indeterminate. The physician may complete this step by announcing clinical decision-making to the team at any time. The nurse will request a decision huddle at 25 minutes into the Code Sepsis event if it has not previously been performed.

- 5) Proceed with next therapeutic and/or diagnostic steps including, for confirmed sepsis patients, immediate initiation of an appropriate antibiotic regimen chosen from a range of options contained in a Code Sepsis antibiotic pack brought to the bedside by a pharmacist on protocol activation. Code Sepsis antibiotic regimens have been selected based on published guidelines and local antibiotic resistance patterns with input from ED clinicians, pharmacists, and infectious disease/antibiotic stewardship personnel.
- 6) If initial huddle pronounced sepsis status as "indeterminate," return to step #4 after additional 20-25 minutes to follow up on additional diagnostic results (e.g. urinalysis, complete blood count
- 7) For antibiotic-treated patients, follow-up by antibiotic stewardship pharmacist active de-escalation or cessation as appropriate.

#### Additional protocol elements/details:

- Code Sepsis team members:
  - ED attending physician +/- ED resident physician or medical student
  - o ED triage nurse
  - ED unit coordinator (i.e. unit secretary)
  - o ED nurses x2
  - o ED patient care technician
  - o ED phlebotomist x1-2
  - o ED pharmacist as available
  - o ED X-ray technician
- Code Sepsis electronic order entry: Code Sepsis order sets for diagnostic evaluation and antibiotic treatment will be constructed and activated at the intervention ED's electronic medical record with the beginning of study Phase #2. Order sets will help speed up diagnostic testing and treatment initiation, aid care standardization, and facilitate Code Sepsis event tracking and data collection.
- Code Sepsis clinical team training: With active support from intervention hospital clinical leadership
  as well as Intermountain's system-wide ED leadership team, the Code Sepsis ED Implementation
  Team will provide clinical staff in the implementation ED with training on the Code Sepsis protocol
  during the months prior to study Phase #2. Primary training will include distribution of instructional
  materials, direct education at clinical staff meetings, targeted in-person education, and in situ
  simulation. Primary training will complete early in study Phase #2, with consolidation training,
  protocol reminders, physician detailing, and targeted clinician reeducation continuing through study
  Phase #3.

## 6. DATA COLLECTION AND VARIABLES

Core analyses will employ data collected during routine clinical care and hospital operations. There will be no direct patient contact for collection of identifiable data or specimens.

#### 6.1 Data Collection

Intermountain's Enterprise Data Warehouse (EDW) is a centrally-managed, well-curated, and accessible database linking system-wide clinical, billing, laboratory, and other data.<sup>31</sup> Eligible patient subjects will be identified by project data managers from EDW data, who will generate a dataset specific to the proposed study by linking EDW data to additional data abstracted from the electronic health record. Manual chart review and direct queries to bedside clinicians will be employed as needed to supplement electronically-available data. This encounter level data will be linked to additional data on hospital characteristics, physician and nurse staffing. Long-term mortality data will be obtained through a preexisting linkage to Utah state death records and/or the federal Social Security Death Index. Encounter data will be linked to data on race, ethnicity, and hospital admissions (admit date, type, diagnoses, and costs) stored in the Utah Population Databank. We will employ a preexisting linkage to Utah State death records and the federal Social Security Death Index for mortality ascertainment.

# 6.2 Anonymous Data Collection For Protocol Development and During Live Code Sepsis Activation

The study team will receive notification of Code Sepsis activations. As part of the study operational process, ED clinical leadership and study personnel will directly observe a convenience sample of these events to anonymously record protocol parameters, including team composition and process completion times. In addition, a convenience sample of intervention hospital patients (<10) with sepsis may be observed during the pre-Code Sepsis implementation phase to understand care processes involved in sepsis care. No identifying information about the patient or clinical team will be recorded.

### 6.3 Active Follow-Up for Patients Undergoing Code Sepsis

Via the electronic medical record, a member of the study team will actively monitor Code Sepsis activation patients every 1-3 days until hospital day #7. There will be no direct patient contact.

### 6.4 Protected Health Information

Protected health information including subject encounter codes, medical record numbers, birthdates, encounter event date and times, address, and social security number will be collected during the electronic query to allow manual chart abstraction and manual review of electronic record for data completion and verification.

### 6.5 Variables/data elements

- Patient medical record number(s)
- Patient encounter ID code
- Hospital/facility
- Date of birth
- Age
- Sex
- Race

- Ethnicity
- Marital status
- Preferred language
- Insurance status/type
- Address/zip code (for determination of residence at a nursing facility or other long-term care facility and estimation of socioeconomic status)
- Social Security Number (to assist matching of encounter data to Social Security Death Index and Utah state death records)
- ED disposition
- Hospital disposition
- Date/time of all events related to ED visit and hospitalization (e.g. ED arrival & departure, hospital admission & discharge)
- Date/time antibiotics administered
- Antibiotic utilization
- APACHE II score
- APACHE IV score
- Acute physiology score
- Charlson index
- Elixhauser index
- SOFA score
- Baseline SOFA score over preceding 10 years
- Source of admission (e.g. home, SNF, LTAC, outside hospital)
- Source of infection
- Clinician infection determination, patient illness severity, sepsis status, and agreement with Code Sepsis activation
- Sepsis presence/absence
- Culture results
- Admission diagnosis
- Mode of arrival to ED
- ED triage data including triage acuity score
- Resident involvement in ED care
- Results of all laboratory testing
- Date/time of all laboratory testing
- ED length of stay
- ED vital signs
- ED medications
- ED interventions/procedures
- Date/time, elapsed time, and type of ED events including provider interaction, room placement, disposition
- Date/time of diagnostic testing, vasopressor initiation and other interventions, and management
- Date/time of interventions
- Date/time of blood or body fluid cultures
- Discharge diagnosis and procedure codes
- Billing diagnosis and procedure codes
- Diagnosis-related group
- Hospital length of stay

- In-hospital mortality
- Long-term mortality (e.g. 30d, 90d and 1y mortality)
- Healthcare charges
- ED patient census
- Number of ED beds
- ED patient flow (including counts of patient arrivals, boarding, and admissions)
- Attending physician ED staffing
- Nurse staffing
- Trauma registration status
- Allergies
- Adverse drug reaction events and date/time
- Code Sepsis team activation (Y/N)
- Code Sepsis activation date/time
- Code Sepsis care process completion date/times
- Code Sepsis team function
- Code Sepsis team composition (by role)
- Code Sepsis process adherence

## 6.6 Data Management

Data analysts and research coordinators will collect data and record it in a custom-designed computer database. Data abstraction from electronic medical records will employ either standardized paper data sheets or a custom-designed interface maintained within Intermountain's secure Research Electronic Data Capture (REDCap) platform.<sup>32</sup> Outside REDCap, all study data will be kept in a protected database on a protected computer. Each subject will be assigned a study identification number, and we will maintain minimal patient identifiers. Data for analysis will use study ID codes for patient subjects. Shared or presented data will be in anonymized or aggregate format such that individual patient subjects cannot be reidentified. Any hard copy case report forms will only include study identification numbers, and will be stored in a locked file cabinet.

## 7. DATA ANALYSIS

## 7.1 Introduction to Quasi-Experimental Analysis

This study will measure the effect of implementing a teambased Code Sepsis protocol for ED sepsis patients by comparing risk-adjusted process and patient-centered outcomes before versus after protocol implementation at a single hospital. Results from simple pre/post analyses, however, may be subject to misinterpretation due to secular trends (changes in the measured outcomes over time not attributable to the study intervention). Analyses of Aim III primary and secondary outcomes will therefore employ quasi-experimental methods to eliminate confounding due to secular trends when estimating the effect of Code Sepsis implementation on outcomes. More complex methods of quasi-experimental analysis includes interrupted time series



Figure 4. Difference-in-differences analysis

and regression discontinuity, but are analogous to the relatively simpler approach called *difference-in-difference analysis* (Figure 4).<sup>33</sup> Difference-in-difference analysis uses multivariable linear regression to compare the adjusted mean door-to-antibiotic time (primary outcome) at the intervention hospital preversus post-implementation of the Code Sepsis protocol using the measured change at non-intervention hospitals to control for pre-/post-intervention changes not attributable to protocol implementation.<sup>34</sup>

$$Y_i = \beta_1 \text{ERA}_i + \beta_2 \text{HOSP} + \beta_3 \text{ERA}_i \times \text{HOSP}_i + \beta_4(Z_i)$$

**Figure 5.** Simplified difference-in-differences equation.  $Y_i$  is the door-to-antibiotic time for patient i, HOSP and ERA are, respectively, indicator variables for care at the intervention hospital or an ED arrival date after Code Sepsis implementation, and Z is a vector of covariates.  $\beta_3$  is the coefficient of interest.

This model tests the difference in intervention ED versus non-intervention EDs' differences in outcome before versus after the Code Sepsis implementation (Figures 4-5). The  $\beta_3$  parameter from the regression model depicted in Figure 5

provides the adjusted difference-in-differences estimate and significance tests for the influence of the Code Sepsis intervention on the outcome of interest.

## 7.2 Multivariable models

Multivariable models will be adjusted for demographic and clinical parameters with known or plausible associations with both door-to-antibiotic time and treatment hospital, presentation before or after Code Sepsis implementation, and/or Code Sepsis activation. Evaluation of secondary outcomes will employ an analogous approach using multivariable linear, Poisson, or logistic regression as appropriate. Repeating the quasi-experimental analysis for the primary and key secondary outcomes after stratification (rather than adjustment) by (1) sex and (2) hypotension present versus absent on ED arrival will allow evaluation of whether these patient characteristics modify the effects of Code Sepsis implementation. In order to measure how the Code Sepsis protocol influences the care of its core target population, we will perform analyses comparing selected outcomes among the subset of patients who have ED triage data suggesting a strong possibility of sepsis. Outcomes to be evaluated in the sensitivity analyses will include door-to-antibiotic time, antibiotic treatment fraction, and antibiotic treatment spectrum.

## 7.3 Sample size/power analysis

Using 2013 to 2017 data from our study hospitals, we estimated conservatively that the intervention ED provides care for 1,650 sepsis patients annually (approximately 4.5 sepsis patients per day) and the

control EDs together care for a total of 2,200 sepsis patients annually (approximately 6 sepsis patients per day). Based on the design and our pilot testing of the Code Sepsis protocol, a very conservative estimate of door-to-antibiotic time for patients who receive antibiotics after evaluation under the Code Sepsis protocol is 50 minutes. By comparison, our preliminary data from 2013 to 2017 indicates current mean (SD) door-to-antibiotic time for ED sepsis patients is 170 (±75) minutes and that only 5% of patients currently receive antibiotics within 1 hour of ED arrival. Assuming (again conservatively) that the Code Sepsis protocol is activated for 30% of sepsis patients treated in the intervention ED during the full implementation phase (study phase #3), we will have 90% power to detect a difference-in-differences change of 16 minutes or more in door-to-antibiotic time associated with Code Sepsis implementation, with the measurement population being all ED sepsis patients. Power calculations employed Monte Carlo simulations, for which technical details are available upon request.

## 8. RISK ASSESSMENT

This study involves a before-and-after analysis of the effects of reorganizing standard ED care for sepsis. Patient care will be studied under two designs for standard sepsis care.

### 8.1 Potential Risks

### 8.1.1 Risk of confidentiality breach

Potential consequences of a breach of confidentiality to the subject could include identify loss of privacy, medicolegal liability, theft, embarrassment, or harassment.

### 8.1.2 Risks for control group patients

Aside from issues discussed above, there are no foreseeable risks for ED patients receiving care at a non-intervention hospital or at the intervention hospital during study phase #1 and #2. Sepsis patients arriving to control hospitals will receive standard care throughout the study.

### 8.1.3. Risks to patients exposed to the Code Sepsis protocol

Patients presenting to the intervention hospital during phases #2 and 3 (run-in implementation and full implementation) will be exposed to and may receive care using the "Code Sepsis" version of standard care. The Code Sepsis protocol is designed to accelerate evaluation, testing, and treatments that the patient would have eventually received under now current standard care. The Code Sepsis intervention is therefore expected to pose no more than minimal risks to ED patients exposed to the protocol, including specifically sepsis patients for whom the Code Sepsis protocol is activated. The potential risks to subjects due to this protocol include:

- 1) Adverse drug reactions or antibiotic-associated infections related to unnecessary or overtreatment antibiotic treatment with prespecified regimens.
- 2) Delay in diagnosis of non-infectious problems due to focus on sepsis or infection related to Code Sepsis activation.
- 3) Delay in care related to resource allocation away from non-Code Sepsis patients without sepsis (bystanders without sepsis).
- 4) For sepsis patients for whom the Code Sepsis protocol is <u>not</u> activated (i.e. bystanders <u>with</u> sepsis), delay in care related to lower index of suspicion for sepsis leading to delayed diagnosis or resource allocation away from these patients.

### 8.2 Alternatives to Participation

There are no alternatives to participation in this pragmatic before/after implementation research study.

## 8.3 Minimization of Risks

Federal regulations at 45 CFR 46.111(a)(1) require that risks to subjects are minimized by using procedures which are consistent with sound research design. We will review the electronic medical record of all Code Sepsis activations for potential adverse effects related to study procedures. This will include review of standardized Code Sepsis documentation incorporated into clinical care as part of the care redesign. While there are no foreseeable effects of data collection on the care of patients who receive standard care at the control hospitals (all study phases) or during the pre-intervention phase at Intermountain Medical Center, monitoring of aggregate data quality will include all hospitals and study phases. As necessary, after consultation with the Independent Safety Monitor, study procedures (including the Code Sepsis protocol) will be adjusted or even halted if important adverse effects are

identified. There are several specific elements of study design inherent in the present protocol that meet this human subject protection requirement.

## 8.3.1 Protections against invasion of privacy or breach of confidentiality

Protection of subject identity and prevention of unintentional release of protected information is of paramount importance to the research team.

- <u>Data storage and transfer</u>: Data will be maintained in password-protected, encrypted research servers, REDCap (a secure, HIPAA-compliant system), or password-protected, encrypted computers. Patient identifiers for prehospital data linkage in Aim I will be provided in secure, encrypted electronic format to Department of Health staff for identification of ambulance patient care reports. Matched records will be returned in secure, encrypted electronic format. All devices will have been approved by Intermountain Healthcare or (during matching of ED data to prehospital data) the Utah Department of Health for use with clinical and research data. Both Intermountain and the State of Utah deploy comprehensive information technology support systems to maintain and regularly update computer systems and maintain physical and electronic safeguards for data management. Any paper case report forms will only include study identification numbers, and will be stored in a locked file cabinet. Datasets used for statistical analyses will be deidentified.
- <u>Data access</u>: Only the PI and the study team will have access to identifying information. All
  individuals with access to identifiable data will have all necessary human subjects training,
  including Good Clinical Practice training as required by NIH policy for applicable study team
  members involved in the clinical trial proposed.
- <u>Training</u>: All study personnel will maintain appropriate training in human subjects research and data protection. The PI, primary mentor, and study staff responsible for study coordination, data collection, and data management of the associated clinical trial will maintain Good Clinical Practice training as per NIH policy (NOT-OD-16-148).

#### 8.3.2 Incidental findings

Data review and analysis will use only data collected as part of routine clinical care and operations. We therefore do not expect identification of incidental findings relevant to patient care.

#### 8.3.3 Protection against medicolegal risk

Data on subjects studied in the proposed aims will be kept confidential in accordance with applicable laws and statues.

### 8.3.4 Optimization of Code Sepsis targeting

Optimization of team activation mechanism during phase #2 of Aim III (intervention run-in and optimization) will help maximize false positive and minimize false negative team activations.

## 8.3.4 Protections against overtreatment and anchoring bias

Physicians and other providers will be educated intensively about the protocol, with particular emphasis on the corresponding concepts that (1) a sepsis team activation does not establish a sepsis diagnosis and (2) that the sepsis prediction tool was specifically not designed to capture all patients with sepsis and that, as a consequence, many patients with sepsis will not trigger a Code Sepsis.

#### 8.3.5 Protections against overtreatment and adverse drug reactions

Part of this redesign of standard care is incorporation of both direct pharmacist involvement in the Code Sepsis team and antibiotic stewardship monitoring of antibiotic-treated Code Sepsis patients to reduce antibiotic overtreatment. Pharmacist involvement will also help minimize the risk of preventable adverse drug or allergic reactions.

## 8.4 Potential Benefits of the Proposed Research to Human Subjects and Others

This study has the potential to generate important findings for patients with sepsis and their treating clinicians, including methods to identify sepsis patients at ED triage or in the prehospital setting. Sepsis patients treated in the intervention ED after implementation of the full Code Sepsis protocol could receive faster evaluation, diagnosis, and treatment initiation, leading to improved patient outcomes. The risks to patient confidentiality and the risks for adverse drug reactions appear substantially less than the potential benefit to sepsis patient subjects and the important knowledge gained about delivery of ED sepsis care.

## 8.5 Importance of the Knowledge to be Gained

Patients with sepsis —a syndrome defined by infection associated with acute organ dysfunction — have high mortality. This syndrome is also common, affecting nearly 3% of ED patients in our data. Early antibiotic initiation improves sepsis outcomes, but many ED patients do not receive timely antibiotics. The overall hypothesis of this phase 2a study is that reorganizing standard ED sepsis care around multidisciplinary "Code Sepsis" teams activated prior to or immediately upon patients' ED arrival will reduce door-to-antibiotic times. Aim III of this proposal will determine whether the Code Sepsis protocol is feasible, safe, and effective at decreasing door-to-antibiotic time. Data from human subjects are also necessary to validate triage- or prehospital-based sepsis prediction models that can be customized by users planning sepsis screening, intensive resource mobilization (as is planned here) for sepsis care, or to aid risk/benefit decisions for sepsis treatments with more than minimal risks (Aim I) and to understand how practice patterns or systems of care may be optimized to accelerate time-dependent treatment while minimizing unintended consequences (Aim II). The no-more-than-minimal risks to subjects from observational research (Aims I and IIA), interviews (Aim IIB), or systematically reorganizing sepsis care to accelerate evaluations and treatments patients would receive anyway under current standard care (Aim III) are acceptable in the context of the important knowledge to be gained to improve care for the common and deadly sepsis syndrome.

## 9. HUMAN SUBJECTS

We will prospectively assess the effect of a system-level intervention on the organization of ED sepsis care using an augmented pre-/post-intervention design. In the post-intervention period, the studied intervention — early activation of ED teams for patients likely to have sepsis — will be adopted as standard care at Intermountain Medical Center. As such, no patients arriving to any ED during the pre-intervention or to a non-intervention control ED will be exposed to the intervention. Conversely, all patients arriving to the Intermountain Medical Center ED in the post-intervention phase will be exposed to the intervention.

## 9.1 Selection of Subjects

Federal regulations at 45 CFR 46(a)(3) require the equitable selection of subjects. All eligible patients will be enrolled. Study exclusion criteria neither unjustly exclude classes of individuals from participation in the research nor unjustly include classes of individuals from participation in the research. Hence, the recruitment of subjects conforms to the principle of distributive justice.

#### 9.2 Waiver of Informed Consent and HIPAA Authorization

To allow analysis of patient outcomes in all patients during both the pre- and post-intervention phases and to facilitate future research through creation of a research registry, we will request a waiver of informed consent and HIPAA authorization based on the following criteria as per 45 CFR 46.116(d) and the HIPAA Privacy Rule.

## 9.2.1 Research and registry involve no more than minimal risk

Acceptance is widespread for protocols using pre-arrival notification to activate ED teams for the treatment of other critical illnesses where time-to-treatment determines outcomes. Since the tested exposure will be incorporated into ED care processes as standard care, and will merely accelerate evaluation, testing, and treatment sepsis patients would receive during current (pre-intervention) standard care, patients will overall experience only the risks associated with standard ED clinical care. Research and registry creation involve no direct contact between the study team and patients, only review of records routinely collected for administration and medical care. For a small number of subjects, there will be anonymized monitoring of ED operations in the form of non-interactive observation of Code Sepsis protocol completion involving collection of anonymous data, which would be standard during implementation of any approach to improving standard ED care.

### 9.2.2 No adverse effects on the rights and welfare of participants

Exposure to standard care in the form of the Code Sepsis protocol and research team abstraction of data routinely collected in the course of clinical care should have no influence on the welfare of study subjects. Analysis and registry storage of data recorded as part of routine clinical care and operations should have no influence on the welfare of study subjects. Because risk is minimal given this design, the waiver of consent and authorization will not adversely affect the rights or welfare of subjects.

# 9.2.3 The research and registry could not practicably be carried out without waiver of informed consent

Given the large number of eligible patient subjects (up to 530,000, including approximately 9,450 patients with sepsis in the primary analysis cohort), the research and registry could not practicably be carried out without the waiver of consent. The sample size for this chart review is large enough that including only those data for which consent could be obtained would prohibit conclusions to be drawn

and would compromise the scientific validity of the study, as a large proportion of the data would be eliminated if obtaining consent were a requirement. Obtaining consent would also preclude rapid initiation of the Code Sepsis protocol and rapid antibiotic initiation. The subjects whose records will be reviewed will not be followed beyond their hospitalization (except for routine use of data on long-term mortality obtained via existing linkages) and would be mostly lost to follow up. The proportion of subjects who have relocated or have passed away will likely be a significant percentage of the subject population, and so the research results would not be meaningful and would lose statistical power if obtaining consent were a requirement.

## 9.2.4 Information on the Code Sepsis protocol and study will be available to all ED patients

We will make available patient information sheets describing the Code Sepsis protocol in the intervention emergency department (e.g. lobby, patient information stations, and on request). It is otherwise not possible to provide patient subjects with information about the study as there is no feasible mechanism by which to notify subjects, attempting to do so would substantially increase the risk of a confidentiality breach, and because the information that is found will have no impact on subjects' clinical care.

## 9.2.5 The minimal necessary amount of protected information will be obtained

Only data necessary for the completion of the study will be collected. The patient ID, encounter ID, social security number, address, and date of birth are necessary to allow data linkage, identification of the specific patient encounter for supplemental data abstraction. Event date/times are necessary for care process and outcome measurement, including calculation of the elapsed time related to various patient management actions include the primary outcome. Identifiers will maintained in the registry to facilitate future research.

#### 9.2.6 All data, including PHI, will be securely guarded from improper disclosure

High-level safeguards will be in place to protect subject identity and confidential data, including in data maintained in the research registry. The study and registry data will be kept on encrypted, passwordprotected computers. These computers are routinely used for storage of patient data and research data including subject identifiers. The data will only be accessible to members of the research team, and all members of the research team have completed Human Subjects Protections and understand the importance of protecting subject privacy and confidentiality. No PHI will be recorded on the CRFs for the study dataset. Protected health information will not be reused or disclosed to any other person or entity, except as required by law, for authorized oversight of the research project, for other research as approved by an IRB, or for other research for which the use or disclosure of protected health information would be permitted by under applicable regulations. Minimal identifiers will be maintained linked to the data. Maintaining minimal identifiers linked to the data is necessary to allow (1) manual abstraction of additional data from the electronic medical record and (2) potential future linkage – with IRB approval -- of the data to additional datasets. No individual subject data will be presented in any presentation, publication or report related to this research. Data will be presented only in anonymized or aggregate or as results of statistical analyses and will not include any individual-level data that could be traced to a particular subject.

## 10. MONITORING AND SAFETY REPORTING

On the basis of established precedents in implementation research, using toolkits supplied by NIH institutes and the University of Washington's CTSA-supported Institute for Translational Health Sciences and in consultation with the Intermountain Institutional Review Board (IRB) and National Institutes of Health (NIH) staff, we believe the proposed clinical trial represents no more than minimal risk to exposed patients. The study will thus be overseen by an Independent Safety Monitor (ISM), a practicing ICU physician with extensive experience performing clinical trials but not affiliated with the current trial.

## 10.1 Potential Risks and Benefits for Participants

- Potential risks: The risk level associated with this study is estimated to be no more than minimal, since the studied intervention prehospital activation of ED-based Code Sepsis teams will be adopted as standard care and is designed to accelerate evaluation, testing, and treatments that the patient would have eventually received under current standard care. While the efficient coordination of therapies is novel and likely to improve care overall, we will monitor for the possibility of effects potentially relevant to faster antibiotic therapy, specifically receipt of antibiotics to which the patient is known to be allergic. This possibility is protected against through inclusion of a pharmacist in the Code Sepsis team. Other risks are also minimal and related to loss of confidentiality of data.
- <u>Potential benefits</u>: The potential benefits to study subjects with sepsis treated in the
  intervention ED after implementation of the full Code Sepsis protocol include faster evaluation,
  diagnosis, and treatment initiation leading to improved patient outcomes.

#### 10.2 Adverse Event and Serious Adverse Event Collection

## 10.2.1 Adverse event

A clinical trial adverse event is any untoward medical event associated with the use of the study procedure, whether or not it is considered related to a drug or study procedure. After Code Sepsis intervention, adverse events related or possibly related to study procedures must be evaluated by the PI. The PI, with assistance from study co-investigators as needed, will assess whether there is a reasonable possibility that the study procedure caused the event, based on the criteria below. Investigators will also consider whether the event is unanticipated or unexplained given the patient's clinical course, previous medical conditions, and concomitant medications. If the severe adverse event is judged to be reportable, as outlined below, then the investigator will report to the ISM and IRB his assessment of the potential relatedness of each adverse event to protocol procedure.

The study uses the following AE attribution scale:

- <u>Definitely Related</u>: The event follows: a) A reasonable, temporal sequence from a study procedure; and b) Cannot be explained by the known characteristics of the patient's clinical state or other therapies; and c) Evaluation of the patient's clinical state indicates to the investigator that the experience is definitely related to study procedures.
- <u>Probably or Possibly Related</u>: The event should be assessed following the same criteria
  for "Definitely Associated". If in the investigator's opinion at least one or more of the
  criteria are not present, then "probably" or "possibly" associated should be selected.
- <u>Probably Not Related</u>: The event occurred while the patient was on the study but can reasonably be explained by the known characteristics of the patient's clinical state or other therapies.

- <u>Definitely Not Related</u>: The event is definitely produced by the patient's clinical state or by other modes of therapy administered to the patient.
- <u>Uncertain Relationship</u>: The event does not meet any of the criteria previously outlined.

#### 10.2.2 Serious Adverse Event (SAE)

An SAE is any AE that results in any of the following outcomes:

- Death
- A life-threatening experience (that is, immediate risk of dying)
- Event requiring prolongation of existing hospitalization. As per http://www.fda.gov/Safety/MedWatch/HowToReport/ucm053087.htm: Report if admission to the hospital or prolongation of hospitalization was a result of the adverse event. Emergency room visits that do not result in admission to the hospital should be evaluated for one of the other serious outcomes (e.g., life-threatening; required intervention to prevent permanent impairment or damage; other serious medically important event).
- Persistent or significant disability/incapacity. As per http://www.fda.gov/Safety/MedWatch/HowToReport/ucm053087.htm: Report if the adverse event resulted in a substantial disruption of a person's ability to conduct normal life functions, i.e., the adverse event resulted in a significant, persistent or permanent change, impairment, damage or disruption in the patient's body function/structure, physical activities and/or quality of life.
- Important medical events that may not result in death, be life-threatening, or require
  hospitalization may be considered serious adverse events when, based upon
  appropriate medical judgment, they may jeopardize the patient and may require
  medical or surgical intervention to prevent one of the outcomes listed in this definition.

#### 10.2.3 Adverse event monitoring

The PI will review potential adverse events monthly for patients for whom the Code Sepsis protocol was activated during the patient's ED visit. The PI will also review within 72 hours of identification any potential anaphylaxis cases occurring within 24 hours of ED antibiotic initiation in Code Sepsis patients. Adverse events will be monitored via review of the medical record for the first 3 days after Code Sepsis activation or until hospital discharge, whichever occurs first, regardless of the investigator's opinion of causation. Thereafter, serious adverse events are not required to be collected unless routine clinical care monitoring or the PI believes that the event was possibly, probably, or definitely to the Code Sepsis protocol.

## 10.3 Adverse Event and Serious Adverse Event Reporting

We emphasize in AE reporting for this study that the intervention under study is an expedited bundling of established elements of clinical care. Study-specific clinical outcomes of sepsis and ED clinical care are exempt from adverse event reporting *unless* the investigator deems the event to be related to the administration of study drug or the conduct of study procedures (or of uncertain relationship). The following are examples of events that will be considered routinely recorded clinical outcomes:

- Death not related to study procedures.
- Adverse drug reaction (excluding anaphylaxis associated with antibiotic administration) not related to study procedures
- Secondary and healthcare associated infections
- Persistent or progressive organ failure

#### Prolonged hospitalization

The PI will report to the ISM within 72 hours of identification all AEs that are serious and possibly, probably, or definitely related to study procedure (or of uncertain relationship) or are unexpected. If the ISM concurs with the PI's assessment, the AE will be reported to the IRB within 7 business days. Other AEs will be reviewed by the PI on a monthly basis and reported in aggregate to the ISM on a quarterly basis. A summary report on all adverse events will be submitted to the IRB during annual recertification as per IRB guidelines. Good Clinical Practice will be followed for conduct of the study.

## 10.4 Interim Analysis

There will be no interim analyses.

## 10.5 Data and Safety Monitoring

Given that this study is using pre-post method to study implementation of a method to deliver clinical standard-of-care therapies in a more efficient, expeditious, and coordinated manner, the safety monitoring plan will be implemented with the use of an *Independent Safety Monitor (ISM)*. The ISM will monitor participant safety, evaluate the progress of the study, review procedures for maintaining the confidentiality of data, and monitor the quality of data collection, management, and analyses. The PI and study personnel will provide all necessary and requested reports to the ISM in a timely manner. The ISM will have full capacity to end the study at her/his discretion if there is an important safety signal, according to a safety monitoring charter that will be finalized in consultation with NIH and the ISM before study launch. Notably, given that the "intervention" in this trial is a non-randomized implementation of a bundle of timely care for sepsis treatment, the safety monitoring plan will focus on monitoring the Code Sepsis activations. The PI will be responsible for ensuring participants' safety and that the study is conducted according to the IRB-approved research plan on a daily basis.

## 10.5.1 Safety Monitoring Procedures

- 1. Since this research examines implementation of a method to deliver clinical standard-of-care therapies in a more efficient, expeditious, and coordinated manner, the foundation for safety monitoring for this study is the routine quality assurance monitoring of the study hospital's Emergency Department. This quality assurance activity includes review of incident reports for clinical adverse events. The ED physician who serves as site medical director and currently has lead responsibility for monitoring of care quality and safety in each study ED. The study team will be in monthly contact via telephone or email with the ED medical director overseeing quality assurance efforts at the intervention hospital to identify potential concerns possibly, probably, or definitely related to Code Sepsis implementation. If necessary, comparisons to control hospital EDs will be performed on the basis of reports from their medical directors.
- 2. Specific to study procedures, all Code Sepsis activations will be individually evaluated. The PI will review all Code Sepsis activations on a monthly basis. AEs will be reported to the ISM in aggregate on a quarterly basis. The PI will report to the ISM within 72 hours of identification all AEs that are serious and possibly, probably, or definitely related to study procedure (or of uncertain relationship) or are unexpected. The ISM and PI together will reach consensus on the ultimate characterization of these possible serious adverse events (SAEs). If disagreement persists after discussion between the ISM and PI, the ISM will make the final decision about the status of the possible SAE. SAEs will be reported to the IRB within 7 business days.
- 3. If required by NIH or other governing bodies, or based on issues observed during trial conduct, we will convene a Data Safety Monitoring Board (DSMB) of clinical experts and members with

expertise in implementation trials with assistance from the Utah Center for Clinical and Translational Science.

## 10.5.2 Enrollment, procedure, regulatory, and data quality monitoring

Our data monitoring plan will include

- 1. Review of accrued data at monthly study team meetings
- 2. Review of data safety and interim data analysis performed by the independent safety monitor
- 3. Semi-annual audits of study materials by the Intermountain PCCM regulatory affairs group
- 4. An annual review performed by the Intermountain Healthcare IRB

Careful monitoring of the data collection, regulatory adherence, data quality, and study procedures will help to protect the safety of study subjects, the quality of data, and the integrity of the study. The PI or study staff will review all data collection on an ongoing basis for data completeness and accuracy as well as protocol compliance. Data verification for key demographic, exposure, and outcome parameters will be performed on an ongoing basis for a random 5% of all Code Sepsis patients. This will occur on the basis of data reabstraction by someone other than the individual who originally collecting the data or by blinded duplicate data entry. The results of the ongoing data review will be incorporated into each review with the ISM. A statement reflecting the results of the ongoing data review will be incorporated into the annual report for the IRB.

## 10.5.3 Frequency of data and safety monitoring

The PI and study team will review data quality and adverse event reports monthly and meet with the ISM quarterly, either in-person or by teleconference call, to review study progress, data quality, and participants' safety. A summary report on all adverse events and data quality will be submitted to the IRB during annual recertification as per IRB guidelines.

### 10.5.4 Independent safety monitor identify and affiliation

The following individual has agreed to serve as the independent safety monitor for the study:

Eliotte Hirshberg, MD, MS

Division of Pulmonary & Critical Care Medicine, Intermountain Medical Center Associate Professor of Medicine, University of Utah School of Medicine

## 10.5.5 Conflict of interest for independent safety monitor

The ISM will have no direct involvement with the study investigators or intervention. The independent safety monitor will sign a Conflict of Interest Statement which includes current affiliations, if any, with pharmaceutical and biotechnology companies (e.g., stockholder, consultant), and any other relationship that could be perceived as a conflict of interest related to the study and/or associated with commercial interests pertinent to study objectives.

### 10.5.6 Independent safety monitor responsibilities

- Review and approve the research protocol and plans for data safety and monitoring;
- Evaluate the progress of the trial, including periodic assessments of data quality and timeliness, recruitment, accrual, participant risk versus benefit, and other factors that can affect study outcome;

- Consider factors external to the study when relevant information becomes available, such as scientific or therapeutic developments that may have an impact on the safety of the participants or the ethics of the trial;
- Review study performance, make recommendations and assist in the resolution of problems reported by the PI;
- Protect the safety of the study participants;
- Make recommendations to the PI concerning continuation, termination or other modifications of the trial based on the observed adverse effects of the treatment under study;
- Ensure the confidentiality of the study data and the results of monitoring; and,
- Assist the IRB by commenting on any concerns related to study conduct, enrollment, sample size, and/or data collection.

## 10.6 Confidentiality During Adverse Event Reporting

AE reports and annual summaries will not include subject- or group-identifiable material. Each report will only include the identification code. Data will be presented in a blinded manner during any open sessions involving the ISM. At meetings with the ISM or in IRB reports, data and discussion are confidential. Participant identities will not be known to the ISM or to the IRB.

## 11. BIBLIOGRAPHY

- 1. Singer M, Deutschman CS, Seymour CW, et al. The third international consensus definitions for sepsis and septic shock (Sepsis-3). JAMA. 2016;315:801–10.
- 2. Gaieski DF, Edwards JM, Kallan MJ, Carr BG. Benchmarking the incidence and mortality of severe sepsis in the United States. Crit Care Med. 2013;41:1167–74.
- 3. Torio CM, Moore BJ. National Inpatient Hospital Costs: The Most Expensive Conditions by Payer, 2013: Statistical Brief #204. Healthcare Cost and Utilization Project. 2016. Available at: https://www.hcup-us.ahrq.gov/reports/statbriefs/sb204-Most-Expensive-Hospital-Conditions.jsp.: Accessed July 6, 2017.
- 4. Kaukonen K-M, Bailey M, Suzuki S, Pilcher D, Bellomo R. Mortality related to severe sepsis and septic shock among critically ill patients in Australia and New Zealand, 2000-2012. JAMA. 2014;311:1308–16.
- 5. Peltan ID, Mitchell KH, Rudd KE, et al. Physician variation in time to antimicrobial treatment for septic patients presenting to the emergency department. Crit Care Med. 2017;45:1011–8.
- 6. Rivers E, Nguyen B, Havstad S, et al. Early goal-directed therapy in the treatment of severe sepsis and septic shock. New Engl J Med. 2001;345:1368–77.
- 7. ProCESS Investigators, Yealy DM, Kellum JA, et al. A randomized trial of protocol-based care for early septic shock. New Engl J Med. 2014;370:1683–93.
- 8. ARISE Investigators, ANZICS Clinical Trials Group, Peake SL, et al. Goal-directed resuscitation for patients with early septic shock. New Engl J Med. 2014;371:1496–506.
- 9. Kumar A, Roberts D, Wood KE, et al. Duration of hypotension before initiation of effective antimicrobial therapy is the critical determinant of survival in human septic shock. Crit Care Med. 2006;34:1589–96.
- 10. Gaieski DF, Mikkelsen ME, Band RA, et al. Impact of time to antibiotics on survival in patients with severe sepsis or septic shock in whom early goal-directed therapy was initiated in the emergency department. Crit Care Med. 2010;38:1045–53.
- 11. Liu VX, Fielding-Singh V, Greene JD, et al. The timing of early antibiotics and hospital mortality in sepsis. Am J Respir Crit Care Med. 2017;196:856–63.
- 12. Seymour CW, New York State Office of Quality and Patient Safety, Prescott HC, et al. Time to treatment and mortality during mandated emergency care for sepsis. New Engl J Med. 2017;376:2235–44.
- 13. Peltan ID, Brown SM, Bledsoe JR, et al. Emergency department door-to-antibiotic time and long-term mortality in sepsis. Chest. 2019.
- 14. Rhodes A, Evans LE, Alhazzani W, et al. Surviving Sepsis Campaign: International guidelines for management of sepsis and septic shock: 2016. Crit Care Med. 2017;45:486–552.
- 15. Levy MM, Evans LE, Rhodes A. The Surviving Sepsis Campaign Bundle: 2018 update. Intensive Care Med. 2018;44:925–8.
- 16. Peltan ID, Mitchell KH, Rudd KE, et al. Prehospital care and emergency department door-to-antibiotic time in sepsis. Ann Am Thorac Soc. 2018;15:1443–50.
- 17. Peltan ID, Bledsoe JR, Oniki TA, et al. ED crowding is associated with delayed antibiotics for sepsis. Ann Emerg Med. 2018.
- 18. MacKenzie EJ, Rivara FP, Jurkovich GJ, et al. A national evaluation of the effect of trauma-center care on mortality. New Engl J Med. 2006;354:366–78.
- 19. Kim SK, Lee SY, Bae HJ, et al. Pre-hospital notification reduced the door-to-needle time for IV tPA in acute ischaemic stroke. Eur J Neurol. 2009;16:1331–5.
- 20. Mosley I, Nicol M, Donnan G, Patrick I, Kerr F, Dewey H. The impact of ambulance practice on

- acute stroke care. Stroke. 2007;38:2765-70.
- 21. Pedersen SH, Galatius S, Hansen PR, et al. Field triage reduces treatment delay and improves long-term clinical outcome in patients with acute ST-segment elevation myocardial infarction treated with primary percutaneous coronary intervention. J Am Coll Cardiol. 2009;54:2296–302.
- 22. Sejersten M, Sillesen M, Hansen PR, et al. Effect on treatment delay of prehospital teletransmission of 12-lead electrocardiogram to a cardiologist for immediate triage and direct referral of patients with ST-segment elevation acute myocardial infarction to primary percutaneous coronary intervention. Am J Cardiol. 2008;101:941–6.
- 23. Seymour CW, Rea TD, Kahn JM, Walkey AJ, Yealy DM, Angus DC. Severe sepsis in pre-hospital emergency care: analysis of incidence, care, and outcome. Am J Respir Crit Care Med. 2012;186:1264–71.
- 24. Wachter RM, Flanders SA, Fee C, Pronovost PJ. Public reporting of antibiotic timing in patients with pneumonia: lessons from a flawed performance measure. Ann Intern Med. 2008;149:29–32.
- 25. Singer M. Antibiotics for sepsis: Does each hour really count, or is it incestuous amplification? Am J Respir Crit Care Med. 2017;196:800–2.
- 26. Klompas M, Calandra T, Singer M. Antibiotics for sepsis Finding the equilibrium. JAMA. 2018;320:1433–4.
- 27. Croskerry P. From mindless to mindful practice--cognitive bias and clinical decision making. New Engl J Med. 2013;368:2445–8.
- 28. Stenehjem E, Hersh AL, Sheng X, et al. Antibiotic use in small community hospitals. Clin Infect Dis. 2016;63:1273–80.
- 29. Call K, Donohue M, Fontaine G, et al. Care Process Model: Emergency Management of Acute Ischemic Stroke. Intermountain Healthcare. 2017. Available at: https://intermountainhealthcare.org/ext/Dcmnt?ncid=520500199.: Accessed October 27, 2018.
- 30. George P, Wisco DR, Gebel J, Uchino K, Newey CR. Nurses are as specific and are earlier in calling in-hospital stroke alerts compared to physicians. J Stroke Cerebrovasc Dis. 2017;26:917–21.
- 31. Clayton PD, Narus SP, Huff SM, et al. Building a comprehensive clinical information system from components: the approach at Intermountain Health Care. Methods Inf Med. 2003;42:1–7.
- 32. Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009;42:377–81.
- 33. Dimick JB, Ryan AM. Methods for evaluating changes in health care policy: the difference-in-differences approach. JAMA. 2014;312:2401–2.
- 34. Peltan ID, Brown CE, Burke AK, Chow EJ, Rowhani-Rahbar A, Crull MR. The July Effect on maternal peripartum complications before and after resident duty hour reform: a population-based retrospective cohort study. Am J Perinatol. Thieme Medical Publishers, 2017;34:818–25.

## APPENDIX A — Eligible IV and IV-equivalent antibiotics

| Antibiotic | Brand/alternative name | Eligible routes |
|------------------------|---------------------------|-----------------|
| Acyclovir | Zovirax | IV |
| Amikacin | Amikin | IV |
| Amphotericin | Amphotec, Ambisome | IV |
| Ampicillin | Principen | IV |
| Ampicillin/sulbactam | Unasyn | IV |
| Anidulafungin | Eraxis | IV |
| Azithromycin | Zithromax, Zmax, Sumamed | IV |
| Aztreonam | Azactam | IV |
| Caspofungin | Cancidas | IV |
| Cefazolin | Ancef | IV |
| Cefdericol | Fetroja | IV |
| Cefepime | Maxipime | IV |
| Cefoperazone | Cefobid | IV |
| Cefotaxime | Claforan | IV |
| Cefotetan | Cefotan | IV |
| Cefoxitin | Mefoxin | IV |
| Ceftaroline | Teflaro | IV |
| Ceftazidime | Fortaz | IV |
| Ceftazidime/avibactam | Avycaz | IV |
| Ceftizoxime | Cefizox | IV |
| Ceftolozane/tazobactam | Zerbaxa, Ceftolozane | IV |
| Ceftriaxone | Rocephin | IV |
| Cefuroxime | Ceftin, Zinacef | IV |
| Chloramphenicol | Chloromycetin | IV |
| Cidofovir | Vistide | IV |
| Ciprofloxacin | Cipro, Ciprobay, Ciproxin | IV |
| Clindamycin | Cleocin | IV |
| Colistin | Colymycin | IV |
| Dalbavancin | Dalvance | IV |
| Daptomycin | Cubicin | IV |
| Delafloxacin | Baxdela | IV |
| Doripenem | Doribax | IV |
| Doxycycline | Doxychel, Vibramycin | IV |
| Eravacycline | Xerava | IV |
| Ertapenem | Invanz | IV |
| Erythromycin | Erythocin, Erythroped | IV |
| Fidaxomycin | Dificid | PO |
| Fluconazole | Diflucan | IV |
| Ganciclovir | Cytovene | IV |
| Gentamicin | Garamycin | IV |
| Imipenem/cilastin | Primaxin | IV |
| Isavuconazole | Cresemba, Isavuconazonium | IV |
| Itraconazole | Sporanox, Onmel | IV |
| Levofloxacin | Levaquin | IV |
| Linezolid | Zyvox | IV |
| Antibiotic | Brand/alternative name | Eligible routes |
|---|---|---|
| Meropenem | Merrem | IV |
| Meropenem/vaborbactam | Vabomere | IV |
| Metronidazole | Flagyl | IV |
| Micafungin | Mycamine | IV |
| Minocycline | Minocin | IV |
| Moxifloxacin | Avelox | IV |
| Nafcillin | Unipen, Nallpen | IV |
| Ofloxacin | Floxin | IV |
| Omadadcycline | Nuzyra, Paratek | IV |
| Oritavancin | Orbactiv | IV |
| Oseltamavir | Tamiflu | PO |
| Oxacillin | Bastocillin | IV |
| Penicillin | Penicillin V, Pencillin G, Pen VK, Bicillin, Veetids, Pentids, Permapen, Pfizerpen, | IV |
| Peramavir | Rapivab | IV |
| Piperacillin/tazobactam | Zosyn | IV |
| Plazomicin | Zemdri | IV |
| Posaconazole | Noxafil | IV |
| Quinuopristin/dalfopristin | Synercid | IV |
| Remdesivir | Veklury | IV |
| Rifampin | Rifadin | IV |
| Telavancin | Vibativ | IV |
| Tetracycline | Achromycin, Tetracyn, Sumycin, Tetrachel | IV |
| Ticarcillin/clavulanate | Timentin | IV |
| Tidezolid | Sivextro | IV |
| Tigecycline | Tygacil | IV |
| Tobramycin | | IV |
| Trimethoprim/sulfamethoxazole | Bactrim, Septra, Sulfatrim | IV |
| Vancomycin | Vancocin | PO |
| Vancomycin | Vancocin | IV |
| Voriconazole | Vfend | IV |
| Zanamivir | Relenza | IV |

# APPENDIX B — "Sepsis mimic" ICD codes

### B.1 Heart failure diagnosis codes<sup>1</sup>

| ICD-9 | ICD-10 | Description |
|---|---|---|
| 398.,91 | 109.81 | Rheumatic heart failure |
| 402.01 | 111.0 | Hypertensive heart disease with heart failure |
| 402.01 | I11.0 | Hypertensive heart disease with heart failure |
| 402.11 | 111.0 | Hypertensive heart disease with heart failure |
| 404.01 | I11.0<br>I13.0 | Hypertensive heart/kidney dz w/heart failure, stage 1-4 CKD or unspec |
| | | · |
| 404.03 | l13.2 | Hypertensive heart/kidney dz w/heart failure, stage 5 CKD or ESRD |
| 404.11 | 113.0 | Hypertensive heart/kidney dz w/heart failure, stage 1-4 CKD or unspec |
| 404.13 | 113.2 | Hypertensive heart/kidney dz w/heart failure, stage 5 CKD or ESRD |
| 404.91 | 113.0 | Hypertensive heart/kidney dz w/heart failure, stage 1-4 CKD or unspec |
| 404.93 | I13.2 | Hypertensive heart/kidney dz w/heart failure, stage 5 CKD or ESRD |
| 428.0 | 150.9 | Heart failure, unspecified |
| 428.1 | 150.1 | Left heart failure |
| 428.20 | 150.20 | Unspecified systolic heart failure |
| 428.21 | 150.21 | Acute systolic heart failure |
| 428.22 | 150.22 | Chronic systolic heart failure |
| 428.23 | 150.23 | Acute on chronic systolic heart failure |
| 428.30 | 150.30 | Unspecified diastolic heart failure |
| 428.31 | 150.31 | Acute diastolic heart failure |
| 428.32 | 150.32 | Chronic diastolic heart failure |
| 428.33 | 150.33 | Acute on chronic diastolic heart failure |
| 428.40 | 150.40 | Unspecified combined systolic and diastolic heart failure |
| 428.41 | 150.41 | Acute combined systolic and diastolic heart failure |
| 428.42 | 150.42 | Chronic combined systolic and diastolic heart failure |
| 428.43 | 150.43 | Acute on chronic combined systolic and diastolic heart failure |
| 428.9 | 150.810 | Right heart failure, unspecified |
| 428.9 | 150.811 | Acute right heart failure |
| 428.9 | 150.812 | Chronic right heart failure |
| 428.9 | 150.813 | Acute on chronic right heart failure |
| 428.9 | 150.814 | Right heart failure due to left heart failure |
| 428.9 | 150.82 | Biventricular heart failure |
| 428.9 | 150.83 | High output heart failure |
| 428.9 | 150.84 | End stage heart failure |
| 428.9 | 150.89 | Other heart failure |
| 428.9 | 150.9 | Heart failure, unspecified |
| Use only if hel | ow is primary di | agnosis and one of above is second diagnosis |
| - | | Dilated cardiomyopathy |
| 425.4<br>425.5 | 142.0<br>142.6 | Alcoholic cardiomyopathy |
| 425.9 | 142.7 | Cardiomyopathy due to drug and external agent |
| 425.9 | 142.8 | Other cardiomyopathy |
| 425.9 | 142.9 | Cardiomyopathy, unspecified |
| 425.8 | 143 | Cardiomyopathy in diseases classified celsewhere |
| 429.83 | I51.81 | Takotsubo cardiomyopathy |

<sup>&</sup>lt;sup>1</sup> Adapted from: Heart Failure CCW Chronic Conditions Algorithm. CMS Chronic Conditions Data Warehouse. 2018. Available at: https://www.ccwdata.org/web/guest/condition-categories.: Accessed

February 13, 2019.

#### B.2 Pulmonary embolism diagnosis codes<sup>1,2</sup>

| ICD-9 | ICD-10 | Description (from ICD-10) |
|---|---|---|
| 415.11 | | latrogenic pulmonary embolism and infarction |
| 415.13 | 126.02 | Saddle embolus of pulmonary artery with acute cor pulmonale |
| 415.19 | 126.09 | Other pulmonary embolism with acute cor pulmonale |
| 415.13 | 126.92 | Saddle embolus of pulmonary artery without acute cor pulmonale |
| 415.19 | 126.99 | Other pulmonary embolism without acute cor pulmonale |
| 673.20 | 088.219 | Thromboembolism in pregnancy, unspecified trimester |
| 673.21 | 083.22 | Thromboembolism in childbirth |
| 673.22 | 088.22 | Thromboembolism in childbirth |
| 673.23 | 083.211 | Thromboembolism in pregnancy, first trimester |
| 673.23 | 083.212 | Thromboembolism in pregnancy, second trimester |
| 673.23 | 083.213 | Thromboembolism in pregnancy, third trimester |
| 673.24 | O83.23 | Thromboembolism in puerperium |

#### Adapted from:

- 1. Aujesky D, Obrosky DS, Stone RA, Auble TE, Perrier A, Cornuz J, Roy P-M, Fine MJ. Derivation and validation of a prognostic model for pulmonary embolism. Am J Respir Crit Care Med 2005;172:1041–1046.
- 2. Wiener RS, Schwartz LM, Woloshin S. Time trends in pulmonary embolism in the United States: evidence of overdiagnosis. Arch Intern Med 2011;171:831–837.

## B.3 Deep vein thrombosis diagnosis codes<sup>1,2</sup>

| ICD-9 | ICD-10 | Description (from ICD-10) |
|---|---|---|
| 451.11 | 180.10 | Phlebitis/thrombophlebitis of unspecified femoral vein |
| 451.11 | 180.11 | Phlebitis/thrombophlebitis of right femoral vein |
| 451.11 | 180.12 | Phlebitis/thrombophlebitis of left femoral vein |
| 451.11 | 180.13 | Phlebitis/thrombophlebitis of bilateral femoral vein |
| 451.19 | 180.201 | Phlebitis/thrombophlebitis of unspecified deep vessels of right lower extremity |
| 451.19 | 180.202 | Phlebitis/thrombophlebitis of unspecified deep vessels of left lower extremity |
| 451.19 | 180.203 | Phlebitis/thrombophlebitis of unspecified deep vessels of bilateral lower extremity |
| 451.19 | 180.209 | Phlebitis/thrombophlebitis of unspecified deep vessels of unspecified lower extremity |
| 451.19 | 180.221 | Phlebitis/thrombophlebitis of right popliteal vein |
| 451.19 | 180.222 | Phlebitis/thrombophlebitis of right popliteal vein |
| 451.19 | 180.223 | Phlebitis/thrombophlebitis of bilateral popliteal vein |
| 451.19 | 180.229 | Phlebitis/thrombophlebitis of unspecified popliteal vein |
| 451.19 | 180.231 | Phlebitis/thrombophlebitis of right tibial vein |
| 451.19 | 180.232 | Phlebitis/thrombophlebitis of right tibial vein |
| 451.19 | 180.233 | Phlebitis/thrombophlebitis of bilateral tibial vein |
| 451.19 | 180.239 | Phlebitis/thrombophlebitis of unspecified tibial vein |
| 451.19 | 180.291 | Phlebitis/thrombophlebitis of other deep vessels of right lower extremity |
| 451.19 | 180.292 | Phlebitis/thrombophlebitis of other deep vessels of left lower extremity |
| 451.19 | 180.293 | Phlebitis/thrombophlebitis of other deep vessels of bilateral lower extremity |
| 451.19 | 180.299 | Phlebitis/thrombophlebitis of other deep vessels of unspecified lower extremity |
| 451.81 | 180.211 | Phlebitis/thrombophlebitis of right iliac vein |
| 451.81 | 180.212 | Phlebitis/thrombophlebitis of left iliac vein |
| 451.81 | 180.213 | Phlebitis/thrombophlebitis of bilateral iliac vein |
| 453.81 | 180.219 | Phlebitis/thrombophlebitis of unspecified iliac vein |
| 451.11 | 180.10 | Phlebitis/thrombophlebitis of unspecified femoral vein |
| 451.11 | 180.11 | Phlebitis/thrombophlebitis of right femoral vein |
| 451.11 | 180.12 | Phlebitis/thrombophlebitis of left femoral vein |
| 451.11 | 180.13 | Phlebitis/thrombophlebitis of bilateral femoral vein |
| 451.19 | 180.201 | Phlebitis/thrombophlebitis of unspecified deep vessels of right lower extremity |
| 451.19 | 180.202 | Phlebitis/thrombophlebitis of unspecified deep vessels of left lower extremity |
| 451.19 | 180.203 | Phlebitis/thrombophlebitis of unspecified deep vessels of bilateral lower extremity |
| 451.19 | 180.209 | Phlebitis/thrombophlebitis of unspecified deep vessels of unspecified lower extremity |
| 451.19 | 180.221 | Phlebitis/thrombophlebitis of right popliteal vein |
| 451.19 | 180.222 | Phlebitis/thrombophlebitis of right popliteal vein |
| 451.19 | 180.223 | Phlebitis/thrombophlebitis of bilateral popliteal vein |
| 451.19 | 180.229 | Phlebitis/thrombophlebitis of unspecified popliteal vein |
| 451.19 | 180.231 | Phlebitis/thrombophlebitis of right tibial vein |
| 451.19 | 180.232 | Phlebitis/thrombophlebitis of right tibial vein |
| 451.19 | 180.233 | Phlebitis/thrombophlebitis of bilateral tibial vein |
| 451.19 | 180.239 | Phlebitis/thrombophlebitis of unspecified tibial vein |
| 451.19 | 180.291 | Phlebitis/thrombophlebitis of other deep vessels of right lower extremity |
| 451.19 | 180.292 | Phlebitis/thrombophlebitis of other deep vessels of left lower extremity |
| 451.19 | 180.293 | Phlebitis/thrombophlebitis of other deep vessels of bilateral lower extremity |
| 451.19 | 180.299 | Phlebitis/thrombophlebitis of other deep vessels of unspecified lower extremity |

| ICD-9 | ICD-10 | Description (from ICD-10) — CONTINUED |
|---|---|---|
| 451.81 | 180.211 | Phlebitis/thrombophlebitis of right iliac vein |
| 451.81 | 180.212 | Phlebitis/thrombophlebitis of left iliac vein |
| 451.81 | 180.213 | Phlebitis/thrombophlebitis of bilateral iliac vein |
| 453.81 | 180.219 | Phlebitis/thrombophlebitis of unspecified iliac vein |
| 451.83 | | Phlebitis/thrombophlebitis of deep vein of upper extremity |
| 453.40 | 182.401 | Acute embolism/thrombosis of unspecified deep veins of right lower extremity |
| 453.40 | 182.402 | Acute embolism/thrombosis of unspecified deep veins of left lower extremity |
| 453.40 | 182.403 | Acute embolism/thrombosis of unspecified deep veins of bilateral lower extremity |
| 453.40 | 182.409 | Acute embolism/thrombosis of unspecified deep veins of unspecified lower extremity |
| 453.40 | 182.491 | Acute embolism/thrombosis of other deep veins of right lower extremity |
| 453.40 | 182.492 | Acute embolism/thrombosis of other deep veins of left lower extremity |
| 453.40 | 182.493 | Acute embolism/thrombosis of other deep veins of bilateral lower extremity |
| 453.40 | 182.499 | Acute embolism/thrombosis of other deep veins of unspecified lower extremity |
| 453.41 | 182.411 | Acute embolism/thrombosis of right femoral vein |
| 453.41 | 182.412 | Acute embolism/thrombosis of left femoral vein |
| 453.41 | 182.413 | Acute embolism/thrombosis of bilateral femoral vein |
| 453.41 | 182.419 | Acute embolism/thrombosis of unspecified femoral vein |
| 453.41 | 182.421 | Acute embolism/thrombosis of right iliac vein |
| 453.41 | 182.422 | Acute embolism/thrombosis of left iliac vein |
| 453.41 | 182.423 | Acute embolism/thrombosis of bilateral iliac vein |
| 453.41 | 182.429 | Acute embolism/thrombosis of unspecified iliac vein |
| 453.41 | 182.4Y1 | Acute embolism/thrombosis of unspecified veins of right proximal lower extremity |
| 453.41 | 182.4Y2 | Acute embolism/thrombosis of unspecified veins of left proximal lower extremity |
| 453.41 | 182.4Y3 | Acute embolism/thrombosis of unspecified veins of bilateral proximal lower extremity |
| 453.41 | 182.4Y9 | Acute embolism/thrombosis of unspecified veins of unspecified prox lower extremity |
| 453.42 | 182.431 | Acute embolism/thrombosis of right popliteal vein |
| 453.42 | 182.432 | Acute embolism/thrombosis of left popliteal vein |
| 453.42 | 182.433 | Acute embolism/thrombosis of bilateral popliteal vein |
| 453.42 | 182.439 | Acute embolism/thrombosis of unspecified popliteal vein |
| 453.42 | 182.441 | Acute embolism/thrombosis of right tibial vein |
| 453.42 | 182.442 | Acute embolism/thrombosis of left tibial vein |
| 453.42 | 182.443 | Acute embolism/thrombosis of bilateral tibial vein |
| 453.42 | 182.449 | Acute embolism/thrombosis of unspecified tibial vein |
| 453.42 | 182.4Z1 | Acute embolism/thrombosis of unspecified veins of right distal lower extremity |
| 453.42 | I82.4Z2 | Acute embolism/thrombosis of unspecified veins of left distal lower extremity |
| 453.42 | I82.4Z3 | Acute embolism/thrombosis of unspecified veins of bilateral distal lower extremity |
| 453.42 | 182.4Z9 | Acute embolism/thrombosis of unspecified veins of unspecified distal lower extremity |
| | 182.621 | Acute embolism/thrombosis of deep veins of right upper extremity |
| | 182.622 | Acute embolism/thrombosis of deep veins of left upper extremity |
| | 182.623 | Acute embolism/thrombosis of deep veins of bilateral upper extremity |
| | 182.629 | Acute embolism/thrombosis of deep veins of unspecified upper extremity |

| ICD-9 | ICD-10 | Description (from ICD-10) — CONTINUED |
|---|---|---|
| 671.30 | 022.30 | Deep phlebothrombosis in pregnancy, unspecified trimester |
| 671.31 | 087.1 | Deep phlebothrombosis in the peurperium |
| 671.33 | 022.31 | Deep phlebothrombosis in pregnancy, first trimester |
| 671.33 | 022.32 | Deep phlebothrombosis in pregnancy, second trimester |
| 671.33 | 022.33 | Deep phlebothrombosis in pregnancy, third trimester |
| 671.40 | 087.1 | Deep phlebothrombosis, postpartum, unspecified as to episode of care |
| 671.42 | 087.1 | Deep phlebothrombosis, postpartum, delivered |
| 671.44 | 087.1 | Deep phlebothrombosis, postpartum, postpartum condition |

#### Adapted from:

- 1. White RH, Garcia M, Sadeghi B, Tancredi DJ, Zrelak P, Cuny J, Sama P, Gammon H, Schmaltz S, Romano PS. Evaluation of the predictive value of ICD-9-CM coded administrative data for venous thromboembolism in the United States. Thromb Res 2010;126:61–67.
- 2. Kniffin WD, Baron JA, Barrett J, Birkmeyer JD, Anderson FA. The epidemiology of diagnosed pulmonary embolism and deep venous thrombosis in the elderly. Arch Intern Med 1994;154:861–866.

## APPENDIX C — Diagnosis codes for adverse drug reaction

Adapted from: Hohl CM, Karpov A, Reddekopp L, Doyle-Waters M, Stausberg J. ICD-10 codes used to

identify adverse drug events in administrative data: a systematic review. J Am Med

Inform Assoc. 2014;21:547–57.

| ICD-10-CM | <b>Anaphylaxis</b> | <u>Description</u> |
|---|---|---|
| A0471 | | Enterocolitis due to Clostridium difficile, recurrent |
| A0472 | | Enterocolitis due to Clostridium difficile, not specified as recurrent |
| D590 | | Drug-induced autoimmune hemolytic anemia |
| D592 | | Drug-induced nonautoimmune hemolytic anemia |
| D7212 | | Drug rash with eosinophilia and systemic symptoms syndrome |
| E064 | | Drug-induced thyroiditis |
| E160 | | Drug-induced hypoglycemia without coma |
| G210 | | Malignant neuroleptic syndrome |
| G2402 | | Drug induced acute dystonia |
| G2409 | | Other drug induced dystonia |
| G251 | | Drug-induced tremor |
| G4440 | | Drug-induced headache, not elsewhere classified, not intractable |
| G4441 | | Drug-induced headache, not elsewhere classified, intractable |
| G620 | | Drug-induced polyneuropathy |
| G720 | | Drug-induced myopathy |
| 1427 | | Cardiomyopathy due to drug and external agent |
| 1952 | | Hypotension due to drugs |
| J702 | | Acute drug-induced interstitial lung disorders |
| J704 | | Drug-induced interstitial lung disorders, unspecified |
| K710 | | Toxic liver disease with cholestasis |
| K7110 | | Toxic liver disease with hepatic necrosis, without coma |
| K7111 | | Toxic liver disease with hepatic necrosis, with coma |
| K712 | | Toxic liver disease with acute hepatitis |
| K716 | | Toxic liver disease with hepatitis, not elsewhere classified |
| K719 | | Toxic liver disease, unspecified |
| K8530 | | Drug induced acute pancreatitis without necrosis or infection |
| K8531 | | Drug induced acute pancreatitis with uninfected necrosis |
| K8532 | | Drug induced acute pancreatitis with infected necrosis |
| L233 | | Allergic contact dermatitis due to drugs in contact with skin |
| L244 | | Irritant contact dermatitis due to drugs in contact with skin |
| L251 | | Unspecified contact dermatitis due to drugs in contact with skin |
| L270 | | Generalized skin eruption due to drugs and medicaments taken internally |
| L271 | | Localized skin eruption due to drugs and medicaments taken internally |
| L278 | | Dermatitis due to other substances taken internally |
| L279 | | Dermatitis due to unspecified substance taken internally |
| L500 | | Allergic urticaria |
| L509 | | Urticaria, unspecified |
| L510 | | Nonbullous erythema multiforme |
| L511 | | Stevens-Johnson syndrome |
| L512 | | Toxic epidermal necrolysis [Lyell] |

| ICD-10-CM | Anaphylaxis | Description |
|---|---|---|
| L513 | | Stevens-Johnson syndrome-toxic epidermal necrolysis overlap syndrome |
| L518 | | Other erythema multiforme |
| L519 | | Erythema multiforme, unspecified |
| L52 | | Erythema nodosum |
| L530 | | Toxic erythema |
| L531 | | Erythema annulare centrifugum |
| N141 | | Nephropathy induced by other drugs, medicaments and biological |
| | | substances |
| N142 | | Nephropathy induced by unspecified drug, medicament or biological |
| | | substance |
| N144 | | Toxic nephropathy, not elsewhere classified |
| R502 | | Drug induced fever |
| T360X1A | | Poisoning by penicillins, accidental (unintentional), initial encounter |
| T360X1D | | Poisoning by penicillins, accidental (unintentional), subsequent encounter |
| T360X1S | | Poisoning by penicillins, accidental (unintentional), sequela |
| T360X4A | | Poisoning by penicillins, undetermined, initial encounter |
| T360X4D | | Poisoning by penicillins, undetermined, subsequent encounter |
| T360X4S | | Poisoning by penicillins, undetermined, sequela |
| T360X5A | | Adverse effect of penicillins, initial encounter |
| T360X5D | | Adverse effect of penicillins, subsequent encounter |
| T360X5S | | Adverse effect of penicillins, sequela |
| T360X6A | | Underdosing of penicillins, initial encounter |
| T360X6D | | Underdosing of penicillins, subsequent encounter |
| T360X6S | | Underdosing of penicillins, sequela |
| T361X1A | | Poisoning by cephalosporins and other beta-lactam antibiotics, accidental |
| | | (unintentional), initial encounter |
| T361X1D | | Poisoning by cephalosporins and other beta-lactam antibiotics, accidental |
| | | (unintentional), subsequent encounter |
| T361X1S | | Poisoning by cephalosporins and other beta-lactam antibiotics, accidental |
| | | (unintentional), sequela |
| T361X4A | | Poisoning by cephalosporins and other beta-lactam antibiotics, |
| | | undetermined, initial encounter |
| T361X4D | | Poisoning by cephalosporins and other beta-lactam antibiotics, |
| | | undetermined, subsequent encounter |
| T361X4S | | Poisoning by cephalosporins and other beta-lactam antibiotics, |
| | | undetermined, sequela |
| T361X5A | | Adverse effect of cephalosporins and other beta-lactam antibiotics, initial |
| | | encounter |
| T361X5D | | Adverse effect of cephalosporins and other beta-lactam antibiotics, |
| | | subsequent encounter |
| T361X5S | | Adverse effect of cephalosporins and other beta-lactam antibiotics, |
| | | sequela |
| T361X6A | | Underdosing of cephalosporins and other beta-lactam antibiotics, initial |
| T0.641/65 | | encounter |
| T361X6D | | Underdosing of cephalosporins and other beta-lactam antibiotics, |
| T2641/66 | | subsequent encounter |
| T361X6S | | Underdosing of cephalosporins and other beta-lactam antibiotics, sequela |

| ICD-10-CM | <u>Anaphylaxis</u> | Description |
|---|---|---|
| T362X1A | · mapy.axio | Poisoning by chloramphenicol group, accidental (unintentional), initial |
| | | encounter |
| T362X1D | | Poisoning by chloramphenicol group, accidental (unintentional), |
| | | subsequent encounter |
| T362X1S | | Poisoning by chloramphenicol group, accidental (unintentional), sequela |
| T362X4A | | Poisoning by chloramphenicol group, undetermined, initial encounter |
| T362X4D | | Poisoning by chloramphenicol group, undetermined, subsequent |
| | | encounter |
| T362X4S | | Poisoning by chloramphenicol group, undetermined, sequela |
| T362X5A | | Adverse effect of chloramphenicol group, initial encounter |
| T362X5D | | Adverse effect of chloramphenicol group, subsequent encounter |
| T362X5S | | Adverse effect of chloramphenicol group, sequela |
| T362X6A | | Underdosing of chloramphenicol group, initial encounter |
| T362X6D | | Underdosing of chloramphenicol group, subsequent encounter |
| T362X6S | | Underdosing of chloramphenicol group, sequela |
| T363X1A | | Poisoning by macrolides, accidental (unintentional), initial encounter |
| T363X1D | | Poisoning by macrolides, accidental (unintentional), subsequent |
| | | encounter |
| T363X1S | | Poisoning by macrolides, accidental (unintentional), sequela |
| T363X4A | | Poisoning by macrolides, undetermined, initial encounter |
| T363X4D | | Poisoning by macrolides, undetermined, subsequent encounter |
| T363X4S | | Poisoning by macrolides, undetermined, sequela |
| T363X5A | | Adverse effect of macrolides, initial encounter |
| T363X5D | | Adverse effect of macrolides, subsequent encounter |
| T363X5S | | Adverse effect of macrolides, sequela |
| T363X6A | | Underdosing of macrolides, initial encounter |
| T363X6D | | Underdosing of macrolides, subsequent encounter |
| T363X6S | | Underdosing of macrolides, sequela |
| T364X1A | | Poisoning by tetracyclines, accidental (unintentional), initial encounter |
| T364X1D | | Poisoning by tetracyclines, accidental (unintentional), subsequent |
| | | encounter |
| T364X1S | | Poisoning by tetracyclines, accidental (unintentional), sequela |
| T364X4A | | Poisoning by tetracyclines, undetermined, initial encounter |
| T364X4D | | Poisoning by tetracyclines, undetermined, subsequent encounter |
| T364X4S | | Poisoning by tetracyclines, undetermined, sequela |
| T364X5A | | Adverse effect of tetracyclines, initial encounter |
| T364X5D | | Adverse effect of tetracyclines, subsequent encounter |
| T364X5S | | Adverse effect of tetracyclines, sequela |
| T364X6A | | Underdosing of tetracyclines, initial encounter |
| T364X6D | | Underdosing of tetracyclines, subsequent encounter |
| T364X6S | | Underdosing of tetracyclines, sequela |
| T365X1A | | Poisoning by aminoglycosides, accidental (unintentional), initial |
| T065145 | | encounter |
| T365X1D | | Poisoning by aminoglycosides, accidental (unintentional), subsequent |
| T067145 | | encounter |
| T365X1S | | Poisoning by aminoglycosides, accidental (unintentional), sequela |
| T365X4A | | Poisoning by aminoglycosides, undetermined, initial encounter |

| ICD-10-CM | <u>Anaphylaxis</u> | Description |
|---|---|---|
| T365X4D | | Poisoning by aminoglycosides, undetermined, subsequent encounter |
| T365X4S | | Poisoning by aminoglycosides, undetermined, sequela |
| T365X5A | | Adverse effect of aminoglycosides, initial encounter |
| T365X5D | | Adverse effect of aminoglycosides, subsequent encounter |
| T365X5S | | Adverse effect of aminoglycosides, sequela |
| T365X6A | | Underdosing of aminoglycosides, initial encounter |
| T365X6D | | Underdosing of aminoglycosides, subsequent encounter |
| T365X6S | | Underdosing of aminoglycosides, sequela |
| T366X1A | | Poisoning by rifampicins, accidental (unintentional), initial encounter |
| T366X1D | | Poisoning by rifampicins, accidental (unintentional), subsequent |
| | | encounter |
| T366X1S | | Poisoning by rifampicins, accidental (unintentional), sequela |
| T366X4A | | Poisoning by rifampicins, undetermined, initial encounter |
| T366X4D | | Poisoning by rifampicins, undetermined, subsequent encounter |
| T366X4S | | Poisoning by rifampicins, undetermined, sequela |
| T366X5A | | Adverse effect of rifampicins, initial encounter |
| T366X5D | | Adverse effect of rifampicins, subsequent encounter |
| T366X5S | | Adverse effect of rifampicins, sequela |
| T366X6A | | Underdosing of rifampicins, initial encounter |
| T366X6D | | Underdosing of rifampicins, subsequent encounter |
| T366X6S | | Underdosing of rifampicins, sequela |
| T367X1A | | Poisoning by antifungal antibiotics, systemically used, accidental (unintentional), initial encounter |
| T367X1D | | Poisoning by antifungal antibiotics, systemically used, accidental |
| | | (unintentional), subsequent encounter |
| T367X1S | | Poisoning by antifungal antibiotics, systemically used, accidental |
| | | (unintentional), sequela |
| T367X4A | | Poisoning by antifungal antibiotics, systemically used, undetermined, initial encounter |
| T367X4D | | Poisoning by antifungal antibiotics, systemically used, undetermined, |
| | | subsequent encounter |
| T367X4S | | Poisoning by antifungal antibiotics, systemically used, undetermined, |
| | | sequela |
| T367X5A | | Adverse effect of antifungal antibiotics, systemically used, initial |
| | | encounter |
| T367X5D | | Adverse effect of antifungal antibiotics, systemically used, subsequent |
| | | encounter |
| T367X5S | | Adverse effect of antifungal antibiotics, systemically used, sequela |
| T367X6A | | Underdosing of antifungal antibiotics, systemically used, initial encounter |
| T367X6D | | Underdosing of antifungal antibiotics, systemically used, subsequent encounter |
| T367X6S | | Underdosing of antifungal antibiotics, systemically used, sequela |
| T368X1A | | Poisoning by other systemic antibiotics, accidental (unintentional), initial |
| ISOUTH | | encounter |
| T368X1D | | Poisoning by other systemic antibiotics, accidental (unintentional), |
| T2C0V4C | | subsequent encounter |
| T368X1S | | Poisoning by other systemic antibiotics, accidental (unintentional), |

| ICD-10-CM | <u>Anaphylaxis</u> | <u>Description</u> |
|---|---|---|
| | | sequela |
| T368X4A | | Poisoning by other systemic antibiotics, undetermined, initial encounter |
| T368X4D | | Poisoning by other systemic antibiotics, undetermined, subsequent |
| | | encounter |
| T368X4S | | Poisoning by other systemic antibiotics, undetermined, sequela |
| T368X5A | | Adverse effect of other systemic antibiotics, initial encounter |
| T368X5D | | Adverse effect of other systemic antibiotics, subsequent encounter |
| T368X5S | | Adverse effect of other systemic antibiotics, sequela |
| T368X6A | | Underdosing of other systemic antibiotics, initial encounter |
| T368X6D | | Underdosing of other systemic antibiotics, subsequent encounter |
| T368X6S | | Underdosing of other systemic antibiotics, sequela |
| T3691XA | | Poisoning by unspecified systemic antibiotic, accidental (unintentional), initial encounter |
| T3691XD | | Poisoning by unspecified systemic antibiotic, accidental (unintentional), subsequent encounter |
| T3691XS | | Poisoning by unspecified systemic antibiotic, accidental (unintentional), sequela |
| T3694XA | | Poisoning by unspecified systemic antibiotic, undetermined, initial encounter |
| T3694XD | | Poisoning by unspecified systemic antibiotic, undetermined, subsequent |
| 1303470 | | encounter |
| T3694XS | | Poisoning by unspecified systemic antibiotic, undetermined, sequela |
| T3695XA | | Adverse effect of unspecified systemic antibiotic, initial encounter |
| T3695XD | | Adverse effect of unspecified systemic antibiotic, subsequent encounter |
| T3695XS | | Adverse effect of unspecified systemic antibiotic, sequela |
| T3696XA | | Underdosing of unspecified systemic antibiotic, initial encounter |
| T3696XD | | Underdosing of unspecified systemic antibiotic, subsequent encounter |
| T3696XS | | Underdosing of unspecified systemic antibiotic, sequela |
| T370X1A | | Poisoning by sulfonamides, accidental (unintentional), initial encounter |
| T370X1D | | Poisoning by sulfonamides, accidental (unintentional), subsequent encounter |
| T370X1S | | Poisoning by sulfonamides, accidental (unintentional), sequela |
| T370X4A | | Poisoning by sulfonamides, undetermined, initial encounter |
| T370X4D | | Poisoning by sulfonamides, undetermined, subsequent encounter |
| T370X4S | | Poisoning by sulfonamides, undetermined, sequela |
| T370X5A | | Adverse effect of sulfonamides, initial encounter |
| T370X5D | | Adverse effect of sulfonamides, subsequent encounter |
| T370X5S | | Adverse effect of sulfonamides, sequela |
| T370X6A | | Underdosing of sulfonamides, initial encounter |
| T370X6D | | Underdosing of sulfonamides, subsequent encounter |
| T370X6S | | Underdosing of sulfonamides, sequela |
| T371X1A | | Poisoning by antimycobacterial drugs, accidental (unintentional), initial |
| | | encounter |
| T371X1D | | Poisoning by antimycobacterial drugs, accidental (unintentional), |
| | | subsequent encounter |
| T371X1S | | Poisoning by antimycobacterial drugs, accidental (unintentional), sequela |
| T371X4A | | Poisoning by antimycobacterial drugs, undetermined, initial encounter |

| ICD-10-CM | <u>Anaphylaxis</u> | Description |
|---|---|---|
| T371X4D | | Poisoning by antimycobacterial drugs, undetermined, subsequent |
| | | encounter |
| T371X4S | | Poisoning by antimycobacterial drugs, undetermined, sequela |
| T371X5A | | Adverse effect of antimycobacterial drugs, initial encounter |
| T371X5D | | Adverse effect of antimycobacterial drugs, subsequent encounter |
| T371X5S | | Adverse effect of antimycobacterial drugs, sequela |
| T371X6A | | Underdosing of antimycobacterial drugs, initial encounter |
| T371X6D | | Underdosing of antimycobacterial drugs, subsequent encounter |
| T371X6S | | Underdosing of antimycobacterial drugs, sequela |
| T372X1A | | Poisoning by antimalarials and drugs acting on other blood protozoa, accidental (unintentional), initial encounter |
| T372X1D | | Poisoning by antimalarials and drugs acting on other blood protozoa, |
| | | accidental (unintentional), subsequent encounter |
| T372X1S | | Poisoning by antimalarials and drugs acting on other blood protozoa, |
| T272V4A | | accidental (unintentional), sequela |
| T372X4A | | Poisoning by antimalarials and drugs acting on other blood protozoa, undetermined, initial encounter |
| T372X4D | | Poisoning by antimalarials and drugs acting on other blood protozoa, |
| | | undetermined, subsequent encounter |
| T372X4S | | Poisoning by antimalarials and drugs acting on other blood protozoa, |
| | | undetermined, sequela |
| T372X5A | | Adverse effect of antimalarials and drugs acting on other blood protozoa, initial encounter |
| T372X5D | | Adverse effect of antimalarials and drugs acting on other blood protozoa, |
| | | subsequent encounter |
| T372X5S | | Adverse effect of antimalarials and drugs acting on other blood protozoa, |
| | | sequela |
| T372X6A | | Underdosing of antimalarials and drugs acting on other blood protozoa, initial encounter |
| T372X6D | | Underdosing of antimalarials and drugs acting on other blood protozoa, |
| | | subsequent encounter |
| T372X6S | | Underdosing of antimalarials and drugs acting on other blood protozoa, |
| | | sequela |
| T373X1A | | Poisoning by other antiprotozoal drugs, accidental (unintentional), initial encounter |
| T373X1D | | Poisoning by other antiprotozoal drugs, accidental (unintentional), |
| | | subsequent encounter |
| T373X1S | | Poisoning by other antiprotozoal drugs, accidental (unintentional), |
| | | sequela |
| T373X4A | | Poisoning by other antiprotozoal drugs, undetermined, initial encounter |
| T373X4D | | Poisoning by other antiprotozoal drugs, undetermined, subsequent encounter |
| T373X4S | | Poisoning by other antiprotozoal drugs, undetermined, sequela |
| T373X5A | | Adverse effect of other antiprotozoal drugs, initial encounter |
| T373X5D | | Adverse effect of other antiprotozoal drugs, subsequent encounter |
| T373X5S | | Adverse effect of other antiprotozoal drugs, sequela |
| T373X6A | | Underdosing of other antiprotozoal drugs, initial encounter |

| ICD-10-CM | Anaphylaxis | Description |
|---|---|---|
| T373X6D | | Underdosing of other antiprotozoal drugs, subsequent encounter |
| T373X6S | | Underdosing of other antiprotozoal drugs, sequela |
| T374X1A | | Poisoning by anthelminthics, accidental (unintentional), initial encounter |
| T374X1D | | Poisoning by anthelminthics, accidental (unintentional), subsequent |
| | | encounter |
| T374X1S | | Poisoning by anthelminthics, accidental (unintentional), sequela |
| T374X4A | | Poisoning by anthelminthics, undetermined, initial encounter |
| T374X4D | | Poisoning by anthelminthics, undetermined, subsequent encounter |
| T374X4S | | Poisoning by anthelminthics, undetermined, sequela |
| T374X5A | | Adverse effect of anthelminthics, initial encounter |
| T374X5D | | Adverse effect of anthelminthics, subsequent encounter |
| T374X5S | | Adverse effect of anthelminthics, sequela |
| T374X6A | | Underdosing of anthelminthics, initial encounter |
| T374X6D | | Underdosing of anthelminthics, subsequent encounter |
| T374X6S | | Underdosing of anthelminthics, sequela |
| T375X1A | | Poisoning by antiviral drugs, accidental (unintentional), initial encounter |
| T375X1D | | Poisoning by antiviral drugs, accidental (unintentional), subsequent encounter |
| T375X1S | | Poisoning by antiviral drugs, accidental (unintentional), sequela |
| T375X4A | | Poisoning by antiviral drugs, undetermined, initial encounter |
| T375X4D | | Poisoning by antiviral drugs, undetermined, subsequent encounter |
| T375X4S | | Poisoning by antiviral drugs, undetermined, sequela |
| T375X5A | | Adverse effect of antiviral drugs, initial encounter |
| T375X5D | | Adverse effect of antiviral drugs, subsequent encounter |
| T375X5S | | Adverse effect of antiviral drugs, sequela |
| T375X6A | | Underdosing of antiviral drugs, initial encounter |
| T375X6D | | Underdosing of antiviral drugs, subsequent encounter |
| T375X6S | | Underdosing of antiviral drugs, sequela |
| T378X1A | | Poisoning by other specified systemic anti-infectives and antiparasitics, |
| | | accidental (unintentional), initial encounter |
| T378X1D | | Poisoning by other specified systemic anti-infectives and antiparasitics, |
| | | accidental (unintentional), subsequent encounter |
| T378X1S | | Poisoning by other specified systemic anti-infectives and antiparasitics, |
| | | accidental (unintentional), sequela |
| T378X4A | | Poisoning by other specified systemic anti-infectives and antiparasitics, |
| | | undetermined, initial encounter |
| T378X4D | | Poisoning by other specified systemic anti-infectives and antiparasitics, |
| | | undetermined, subsequent encounter |
| T378X4S | | Poisoning by other specified systemic anti-infectives and antiparasitics, |
| | | undetermined, sequela |
| T378X5A | | Adverse effect of other specified systemic anti-infectives and |
| | | antiparasitics, initial encounter |
| T378X5D | | Adverse effect of other specified systemic anti-infectives and |
| | | antiparasitics, subsequent encounter |
| T378X5S | | Adverse effect of other specified systemic anti-infectives and |
| | | antiparasitics, sequela |
| T378X6A | | Underdosing of other specified systemic anti-infectives and antiparasitics, |

| ICD-10-CM Anaphylaxis | |
|---|---|
| T378X6D | initial encounter Underdosing of other specified systemic anti-infectives and antiparasitics, |
| T378X6S | subsequent encounter Underdosing of other specified systemic anti-infectives and antiparasitics, sequela |
| T3791XA | Poisoning by unspecified systemic anti-infective and antiparasitics, accidental (unintentional), initial encounter |
| T3791XD | Poisoning by unspecified systemic anti-infective and antiparasitics, accidental (unintentional), subsequent encounter |
| T3791XS | Poisoning by unspecified systemic anti-infective and antiparasitics, accidental (unintentional), sequela |
| T3794XA | Poisoning by unspecified systemic anti-infective and antiparasitics, undetermined, initial encounter |
| T3794XD | Poisoning by unspecified systemic anti-infective and antiparasitics, undetermined, subsequent encounter |
| T3794XS | Poisoning by unspecified systemic anti-infective and antiparasitics, undetermined, sequela |
| T3795XA | Adverse effect of unspecified systemic anti-infective and antiparasitic, initial encounter |
| T3795XD | Adverse effect of unspecified systemic anti-infective and antiparasitic, subsequent encounter |
| T3795XS | Adverse effect of unspecified systemic anti-infective and antiparasitic, sequela |
| T3796XA | Underdosing of unspecified systemic anti-infectives and antiparasitics, initial encounter |
| T3796XD | Underdosing of unspecified systemic anti-infectives and antiparasitics, subsequent encounter |
| T3796XS | Underdosing of unspecified systemic anti-infectives and antiparasitics, sequela |
| T431X5A | Adverse effect of monoamine-oxidase-inhibitor antidepressants, initial encounter |
| T431X5D | Adverse effect of monoamine-oxidase-inhibitor antidepressants, subsequent encounter |
| T431X5S | Adverse effect of monoamine-oxidase-inhibitor antidepressants, sequela |
| T43215A | Adverse effect of selective serotonin and norepinephrine reuptake inhibitors, initial encounter |
| T43215D | Adverse effect of selective serotonin and norepinephrine reuptake inhibitors, subsequent encounter |
| T43215S | Adverse effect of selective serotonin and norepinephrine reuptake inhibitors, sequela |
| T43225A | Adverse effect of selective serotonin reuptake inhibitors, initial encounter |
| T43225D | Adverse effect of selective serotonin reuptake inhibitors, subsequent encounter |
| T43225S | Adverse effect of selective serotonin reuptake inhibitors, sequela |
| T50901A | Poisoning by unspecified drugs, medicaments and biological substances, accidental (unintentional), initial encounter |
| T50901D | Poisoning by unspecified drugs, medicaments and biological substances, |

| <u>ICD-10-CM</u> | <u>Anaphylaxis</u> | <u>Description</u> |
|---|---|---|
| TE00016 | | accidental (unintentional), subsequent encounter |
| T50901S | | Poisoning by unspecified drugs, medicaments and biological substances, accidental (unintentional), sequela |
| T50904A | | Poisoning by unspecified drugs, medicaments and biological substances, |
| | | undetermined, initial encounter |
| T50904D | | Poisoning by unspecified drugs, medicaments and biological substances, |
| T50904S | | undetermined, subsequent encounter Poisoning by unspecified drugs, medicaments and biological substances, |
| 1309043 | | undetermined, sequela |
| T50905A | | Adverse effect of unspecified drugs, medicaments and biological |
| | | substances, initial encounter |
| T50905D | | Adverse effect of unspecified drugs, medicaments and biological |
| | | substances, subsequent encounter |
| T50905S | | Adverse effect of unspecified drugs, medicaments and biological |
| T50906A | | substances, sequela Underdosing of unspecified drugs, medicaments and biological |
| 130300A | | substances, initial encounter |
| T50906D | | Underdosing of unspecified drugs, medicaments and biological |
| | | substances, subsequent encounter |
| T50906S | | Underdosing of unspecified drugs, medicaments and biological |
| TE0001 A | | substances, sequela |
| T50991A | | Poisoning by other drugs, medicaments and biological substances, accidental (unintentional), initial encounter |
| T50991D | | Poisoning by other drugs, medicaments and biological substances, |
| | | accidental (unintentional), subsequent encounter |
| T50991S | | Poisoning by other drugs, medicaments and biological substances, |
| | | accidental (unintentional), sequela |
| T50994A | | Poisoning by other drugs, medicaments and biological substances, |
| T50994D | | undetermined, initial encounter Poisoning by other drugs, medicaments and biological substances, |
| 1303340 | | undetermined, subsequent encounter |
| T50994S | | Poisoning by other drugs, medicaments and biological substances, |
| | | undetermined, sequela |
| T50995A | | Adverse effect of other drugs, medicaments and biological substances, |
| TEOOOED | | initial encounter |
| T50995D | | Adverse effect of other drugs, medicaments and biological substances, subsequent encounter |
| T50995S | | Adverse effect of other drugs, medicaments and biological substances, |
| | | sequela |
| T50996A | | Underdosing of other drugs, medicaments and biological substances, |
| | | initial encounter |
| T50996D | | Underdosing of other drugs, medicaments and biological substances, |
| T50996S | | subsequent encounter Underdosing of other drugs, medicaments and biological substances, |
| 1303303 | | sequela |
| T782XXA | Χ | Anaphylactic shock, unspecified, initial encounter |
| T782XXD | Χ | Anaphylactic shock, unspecified, subsequent encounter |

| ICD-10-CM | <u>Anaphylaxis</u> | <u>Description</u> |
|---|---|---|
| T782XXS | Χ | Anaphylactic shock, unspecified, sequela |
| T783XXA | Χ | Angioneurotic edema, initial encounter |
| T783XXD | Χ | Angioneurotic edema, subsequent encounter |
| T783XXS | Χ | Angioneurotic edema, sequela |
| T7840XA | | Allergy, unspecified, initial encounter |
| T7840XD | | Allergy, unspecified, subsequent encounter |
| T7840XS | | Allergy, unspecified, sequela |
| T7841XA | | Arthus phenomenon, initial encounter |
| T7841XD | | Arthus phenomenon, subsequent encounter |
| T7841XS | | Arthus phenomenon, sequela |
| T7849XA | | Other allergy, initial encounter |
| T7849XD | | Other allergy, subsequent encounter |
| T7849XS<br>T788XXA | | Other allergy, sequela |
| T788XXD | | Other adverse effects, not elsewhere classified, initial encounter Other adverse effects, not elsewhere classified, subsequent encounter |
| T788XXS | | Other adverse effects, not elsewhere classified, sequela |
| T8051XA | Χ | Anaphylactic reaction due to administration of blood and blood products, |
| 10031/1/( | ^ | initial encounter |
| T8051XD | Х | Anaphylactic reaction due to administration of blood and blood products, |
| | , | subsequent encounter |
| T8051XS | Χ | Anaphylactic reaction due to administration of blood and blood products, |
| | | sequela |
| T8052XA | Χ | Anaphylactic reaction due to vaccination, initial encounter |
| T8052XD | Χ | Anaphylactic reaction due to vaccination, subsequent encounter |
| T8052XS | Χ | Anaphylactic reaction due to vaccination, sequela |
| T8059XA | Χ | Anaphylactic reaction due to other serum, initial encounter |
| T8059XD | Χ | Anaphylactic reaction due to other serum, subsequent encounter |
| T8059XS | Χ | Anaphylactic reaction due to other serum, sequela |
| T8089XA | | Other complications following infusion, transfusion and therapeutic |
| | | injection, initial encounter |
| T8089XD | | Other complications following infusion, transfusion and therapeutic |
| | | injection, subsequent encounter |
| T8089XS | | Other complications following infusion, transfusion and therapeutic |
| | | injection, sequela |
| T8090XA | | Unspecified complication following infusion and therapeutic injection, |
| | | initial encounter |
| T8090XD | | Unspecified complication following infusion and therapeutic injection, |
| T0000V6 | | subsequent encounter |
| T8090XS | | Unspecified complication following infusion and therapeutic injection, |
| TOOCYVA | V | sequela |
| T886XXA | Χ | Anaphylactic reaction due to adverse effect of correct drug or |
| T886XXD | Χ | medicament properly administered, initial encounter Anaphylactic reaction due to adverse effect of correct drug or |
| ΙΟΟΟΛΛΟ | ^ | medicament properly administered, subsequent encounter |
| T886XXS | Χ | Anaphylactic reaction due to adverse effect of correct drug or |
| 1000773 | ^ | medicament properly administered, sequela |
| | | medicament property duministered, sequeia |

| ICD-10-CM | <b>Anaphylaxis</b> | <u>Description</u> |
|---|---|---|
| T887XXA | | Unspecified adverse effect of drug or medicament, initial encounter |
| T888XXA | | Other specified complications of surgical and medical care, not elsewhere |
| | | classified, initial encounter |
| T889XXA | | Complication of surgical and medical care, unspecified, initial encounter |
| Y631 | | Incorrect dilution of fluid used during infusion |
| Y638 | | Failure in dosage during other surgical and medical care |
| Y639 | | Failure in dosage during unspecified surgical and medical care |
| Y640 | | Contaminated medical or biological substance, transfused or infused |
| Y641 | | Contaminated medical or biological substance, injected or used for |
| | | immunization |
| Y651 | | Wrong fluid used in infusion |
| Y66 | | Nonadministration of surgical and medical care |
| Y69 | | Unspecified misadventure during surgical and medical care |